#### The GlaxoSmithKline group of companies

| Division | : | Worldwide Development |
|------------------|---|-----------------------------------|
| Information Type | : | Reporting and Analysis Plan (RAP) |

| Title | : | Reporting and Analysis Plan for BEL116027 A Phase IV,<br>Open-label, Non-randomized, 52-Week Study to Evaluate<br>Treatment Holidays and Rebound Phenomenon After<br>Treatment with Belimumab 10 mg/kg in Systemic Lupus<br>Erythematosus Subjects |
|---|---|---|
| <b>Compound Number</b> | : | GSK1550188 |
| <b>Effective Date</b> | : | 30-JAN-2019 |

## **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol BEL116027.
- This RAP is intended to describe the final analyses required for the study.
- This RAP will be provided to the study team members to convey the content of the Statistical Analysis Complete deliverable.

## **RAP Author(s):**

| Approver | | Date | Approval Method |
|--------------|--------------------|-------------|-----------------|
| Director, Cl | inical Statistics | 29-Jan-2019 | email |
| Director, Cr | illical Statistics | | |

Copyright 2019 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

## The GlaxoSmithKline group of companies

## **RAP Team Approvals:**

| Approver | Date | Approval Method |
|---|---|---|
| Manager, Immuno-Inflammation, Clinical Programming | 28-Jan-2019 | email |
| Senior Director, Immuno-Inflammation,<br>Clinical Development | 28-Jan-2019 | email |
| Manager, Immuno-Inflammation, Clinical Data Management | 28-Jan-2019 | email |
| Clinical Development Manager, Immuno-<br>Inflammation, PCPS | 18-Jan-2019 | email |
| Medical Writing Director, Immuno-<br>Inflammation, Clinical Development | 24-Jan-2019 | email |
| PPD Director, CPMS | 22-Jan -2019 | email |
| SERM Director, II, GCSP | 24-Jan -2019 | email |

## The GlaxoSmithKline group of companies

## **Clinical Statistics and Clinical Programming Line Approvals:**

| Approver | Date | Approval Method |
|---|---|---|
| Line Manager, Immuno-Inflammation, Clinical Programming | 30-Jan-2019 | Pharma TMF<br>eSignature |
| Senior Director, Immuno-Inflammation, Clinical Statistics On behalf of PPD (Line Manager, Immuno-Inflammation, Clinical Statistics) | 30-Jan-2019 | Pharma TMF<br>eSignature |

.

## **TABLE OF CONTENTS**

| | | | PAGE |
|---|---|---|---|
| 1. | INTR | ODUCTION | 9 |
| 2. | VEV I | PROTOCOL INFORMATION | 0 |
| ۷. | 2.1. | | |
| | 2.1.<br>2.2. | Changes to the Protocol Defined Statistical Analysis Plan | |
| | | Study Objective(s) and Endpoint(s) | |
| | 2.3. | Study Design | |
| | 2.4. | Statistical Hypotheses / Statistical Analyses | 14 |
| 3. | PLAN | NED ANALYSES | 15 |
| | 3.1. | Interim Analyses | 15 |
| | 3.2. | Final Analyses | 15 |
| 4. | ANAI | YSIS POPULATIONS | 16 |
| •• | 4.1. | Protocol Deviations | |
| | 7.1. | 1 Totogol Deviations | |
| 5. | | SIDERATIONS FOR DATA ANALYSES AND DATA HANDLING | |
| | | VENTIONS | |
| | 5.1. | Study Treatment Descriptors | |
| | 5.2. | Parent Studies | |
| | 5.3. | Baseline Definitions | |
| | | 5.3.1. Baseline Definitions <sup>1</sup> | |
| | | 5.3.2. Derivations and Handling of Missing Baseline Data | |
| | 5.4. | Multicentre Studies | 19 |
| | 5.5. | Other Considerations for Data Analyses and Data Handling | 00 |
| | | Conventions | 20 |
| 6. | STUE | DY POPULATION ANALYSES | 21 |
| | 6.1. | Overview of Planned Demography, Baseline Characteristics and | |
| | | Medical History Analyses | 21 |
| | 6.2. | Baseline Disease Activity and Other Baseline Endpoints | 21 |
| | 6.3. | Study Population Data for Maintenance Phase Subject Profile | |
| | | • | |
| 7. | | CACY ANALYSES | |
| | 7.1. | Primary Efficacy Analyses | |
| | | 7.1.1. Endpoint / Variables | |
| | | 7.1.2. Summary Measure | |
| | | 7.1.3. Population of Interest | |
| | | 7.1.4. Strategy for Intercurrent (Post-Randomization) Events | 25 |
| | | 7.1.5. Statistical Analyses / Methods | 26 |
| | 7.2. | Secondary Efficacy Analyses | 26 |
| | | 7.2.1. Endpoint / Variables | <mark>26</mark> |
| | | 7.2.1.1. Rate of Flares | <mark>26</mark> |
| | | 7.2.1.2. First Severe SFI Flare | <mark>26</mark> |
| | | 7.2.1.3. Rebound | |
| | | 7.2.1.4. SELENA SLEDAI Scores | <mark>26</mark> |
| | | 7.2.2. Summary Measure | <mark>27</mark> |
| | | 7.2.2.1. Rate of Flares | |
| | | 7.2.2.2. First Severe SFI Flare | <mark>27</mark> |

| | | | 7.2.2.3.<br>7.2.2.4. | | LEDAI Scores | |
|---|---|---|---|---|---|---|
| | | 7 2 2 | 7.2.2.5. | | Corticosteroid Use | |
| | | 7.2.3. | | | ot (Doot Dondoninstian) Frants | |
| | | 7.2.4. | | | nt (Post-Randomization) Events | |
| | | | 7.2.4.1. | | res and First Severe SFI Flare | |
| | | | 7.2.4.2. | | nd SELENA SLEDAI Scores | |
| | | | 7.2.4.3. | | Corticosteroid Use | 28 |
| | | | | 7.2.4.3.1. | Number of days of daily | |
| | | | | | prednisone dose ≥7.5 mg/day | |
| | | | | | and/or increased by 25% | 28 |
| | | | | 7.2.4.3.2. | Number of days of daily | |
| | | | | | prednisone dose ≤7.5 mg/day | |
| | | | | | and/or decreased by 25% | 28 |
| | | 7.2.5. | Statistical | Analyses / N | Nethods | 28 |
| | 7.3. | Explorat | ory Efficacy | / Analyses | | 29 |
| | | 7.3.1. | | | | |
| | | | 7.3.1.1. | | Global Assessment (PGA) | |
| | | | 7.3.1.2. | | , | |
| | | | 7.3.1.3. | | ) | |
| | | 7.3.2. | | | | |
| | | 7.0.2. | 7.3.2.1. | | Global Assessment (PGA) and | |
| | | | 7.0.2.1. | | | 29 |
| | | | 7.3.2.2. | | PS | |
| | | 7.3.3. | | | | |
| | | 7.3.4. | | | nt (Post-Randomization) Events | |
| | | 7.3.4. | 7.3.4.1. | | | |
| | | | 7.3.4.1.<br>7.3.4.2. | • | Global Assessment (PGA) | |
| | | | _ | | | |
| | | 7.3.5. | 7.3.4.3. | | Aothodo | |
| | 7.4 | | | | Methods | |
| | 7.4. | Efficacy | Data for Ma | amtenance P | hase Subject Profile | 30 |
| 0 | CAFE | T\/ | VOEC | | | 24 |
| 8. | | | | | | |
| | 8.1. | | | | | |
| | 8.2. | | | | est Analyses | |
| | | 8.2.1. | • | | | |
| | | | 8.2.1.1. | | ents of Special Interest | |
| | | | 8.2.1.2. | | on systemic reactions by infusion | |
| | | 8.2.2. | | | | |
| | | | 8.2.2.1. | | rents of Special Interest | |
| | | | 8.2.2.2. | | on systemic reactions by infusion | |
| | | 8.2.3. | | | | |
| | | 8.2.4. | Strategy f | or Intercurre | nt (Post-Randomization) Events | 33 |
| | | 8.2.5. | Statistical | Analyses / N | Nethods | 33 |
| | 8.3. | Clinical I | Laboratory | Analyses | | 33 |
| | | 8.3.1. | | | | |
| | | | 8.3.1.1. | | ooratory Results | |
| | | | 8.3.1.2. | | oratory Toxicity Grades | |
| | | | 8.3.1.3. | | oratory Reference Range Shifts | |
| | | | 8.3.1.4. | | bulin Results Relative to the Lower | |
| | | | J.J | | mal | 35 |
| | | 8.3.2. | Summary | | | |
| | | J.J | Jannary | | | |

| | | | 8.3.2.1. | Clinical Laboratory Results | 35 |
|---|---|---|---|---|---|
| | | | 8.3.2.2. | Clinical Laboratory Toxicity Grades | 35 |
| | | | 8.3.2.3. | Clinical Laboratory Reference Range Shifts | |
| | | | 8.3.2.4. | Immunoglobulin Results Relative to the Lower | |
| | | | | Limit of Normal | 35 |
| | | 8.3.3. | Population | of Interest | |
| | | 8.3.4. | | or Intercurrent (Post-Randomization) Events | |
| | | 8.3.5. | | Analyses / Methods | |
| | 8.4. | | | ses | |
| | 0. 1. | 8.4.1. | | Variables | |
| | | 0. 1. 1. | 8.4.1.1. | Immunogenicity | |
| | | | 8.4.1.2. | Vital signs | |
| | | 8.4.2. | - | Measure | |
| | | 0.4.2. | 8.4.2.1. | | |
| | | | 8.4.2.2. | Vital signs | |
| | | 8.4.3. | - | of Interest | |
| | | 8.4.4. | | or Interest:or Interest:or Interest:or Interest: | |
| | | 0.4.4. | 8.4.4.1. | Immunogenicity | |
| | | | 8.4.4.1. | | |
| | | 8.4.5. | • | Vital signs | |
| | 0.5 | | | Analyses / Methods | |
| | 8.5. | Salety D | ata ioi iviali | ntenance Phase Subject Profile | 30 |
| 9. | PHΔR | ΜΔΟΟΚΙΝ | JETIC ANA | LYSES | 30 |
| ٥. | 9.1. | | | inetic Analyses | |
| | 9.1. | 9.1.1. | | Variables | |
| | | 9.1.1. | | Measure | |
| | | 9.1.2. | | | |
| | | | | of Interest | |
| | | 9.1.4.<br>9.1.5. | Statistical | or Intercurrent (Post-Randomization) Events<br>Analyses / Methods | აყ |
| | | 9.1.5. | Statistical | Analyses / Methods | 39 |
| 10 | POPU | I ATION F | PHARMACO | OKINETIC (POPPK) ANALYSES | 40 |
| 10. | 1 01 0 | L/ (1101 <b>1</b> 1 | 11/11/11/11/10 | 51(114E116 (1 61 1 14) / 114/1E16E6 | 40 |
| 11. | BIOMA | ARKER AI | NALYSES. | | 41 |
| | 11.1. | | | Analyses | |
| | | | | Variables | |
| | | | | Measure | |
| | | | 11 1 2 1 | B-Cells | 41 |
| | | | | Autoantibodies, Immunoglobulins and | |
| | | | | Complement | 41 |
| | | | 11.1.2.3. | BLyS Protein | 41 |
| | | 11.1.3. | | of Interest | 41 |
| | | 11.1.4. | | or Intercurrent (Post-Randomization) Events | |
| | | 11.1.5. | | Analyses / Methods | |
| | 11.2. | | er Data for | Maintenance Phase Subjects | 42 |
| | 11.2. | Diomank | or Data for | Maintenance i nase subjects | 42 |
| 12. | REFE | RENCES. | | | 43 |
| | <b></b> | | | | |
| 13. | APPE | NDICES | | | 44 |
| | 13.1. | | | ol Deviation | |
| | 13.2. | | | lle of Activities | |
| | | | | Defined Schedule of Events | |
| | | | | Events Table (Year 1) | |
| | | | | , | _ |

| 13.3. | 13.2.3.<br>Appendi | ix 3: Assessment Windows | |
|---|---|---|---|
| | 13.3.1. | Mapping of the Maintenance Phase Visits for Subjects with an Escape Visit | 50 |
| | 13.3.2. | Mapping of Week 16 and 6-month Follow-up Visits | |
| | 13.3.3. | Analysis Visit and Analysis Visit Number | |
| | 13.3.4. | Windows for Assessment of Post-injection/infusion | |
| | | sensitivity reactions (PISR) and hypersensitivity reactions | |
| | | (HSR) | 52 |
| 13.4. | | ix 4: Study Phases and Treatment Emergent Adverse | |
| | 13.4.1. | | |
| | | 13.4.1.1. Treatment Holiday Group | |
| | | 13.4.1.2. Treatment Control Group | |
| | | 13.4.1.3. Long-term Discontinuation Group | 56 |
| 13.5. | Appendi | ix 5: Data Display Standards & Handling Conventions | |
| | 13.5.1. | Reporting Process | |
| | 13.5.2. | | |
| | 13.5.3. | Reporting Standards for Pharmacokinetic | |
| 13.6. | Appendi | ix 6: Derived and Transformed Data | 60 |
| | 13.6.1. | General | 60 |
| | 13.6.2. | Study Population | |
| | 13.6.3. | Efficacy | 63 |
| | 13.6.4. | Safety | 70 |
| | 13.6.5. | Pharmacokinetic | |
| | 13.6.6. | Biomarker | 72 |
| | | 13.6.6.1. Autoantibody, Complement, Immunoglobulins, | |
| | | and BLyS Protein | |
| 40.7 | Δ | 13.6.6.2. B-cell Subsets | |
| 13.7. | Appendi | ix 7: Reporting Standards for Missing Data | |
| | 13.7.1. | | |
| | 13.7.2. | 3 3 | |
| | 1070 | 13.7.2.1. Handling of Missing and Partial Dates | // |
| | 13.7.3. | Handling of Prohibited Medications, Withdrawals and Deaths | 78 |
| 13.8. | Appendi | ix 8: Values of Potential Clinical Importance | <mark>7</mark> 9 |
| | 13.8.1. | Laboratory Values | |
| | 13.8.2. | Adverse Event and Laboratory Value Severity Grade | |
| | | Tables | |
| 13.9. | | ix 9: Adverse Events of Special Interest | |
| | 13.9.1. | Malignant neoplasms | |
| | 13.9.2. | Post-infusion systemic reactions | |
| | 13.9.3. | Infections | |
| | 4004 | 13.9.3.1. Opportunistic Infections | |
| | 13.9.4. | Mycobacterium Tuberculosis | |
| | 13.9.5. | Herpes Zoster | |
| | 13.9.6. | Pneumonia | |
| | 13.9.7. | Sepsis | |
| | 13.9.8. | Depression/suicide/self-injury | |
| | | 13.9.8.1. Depression (excluding suicide and self-injury) | |
| | 13.9.9. | 13.9.8.2. Suicide and Self-InjuryFatalities | |
| | 13.3.3. | - เ | కర |

| | 13.9.10. | GSK SRT Adjudication of Adverse Events of Special | |
|---|---|---|---|
| | | Interest | |
| | | 13.9.10.1. Malignancies | 93 |
| | | 13.9.10.2. Serious hypersensitivity and post-infusion | |
| | | systemic reactions | 94 |
| | | 13.9.10.3. Potential opportunistic infections | 94 |
| | | 13.9.10.4. Suicide/self-injury | 96 |
| | | 13.9.10.5. Fatalities | 96 |
| 13.10. | Appendix | c 10: Abbreviations & Trade Marks | 97 |
| | 13.10.1. | Abbreviations | 97 |
| | 13.10.2. | Trademarks | 98 |
| 13.11. | Appendix | 11: List of Data Displays | 99 |
| | 13.11.1. | Data Display Numbering | 99 |
| | | Deliverables | |
| | 13.11.3. | Study Population Tables | 100 |
| | 13.11.4. | Study Population Figures | 101 |
| | 13.11.5. | Efficacy Tables | 102 |
| | 13.11.6. | Efficacy Figures | 103 |
| | 13.11.7. | Safety Tables | 104 |
| | 13.11.8. | Safety Figures | 110 |
| | 13.11.9. | Pharmacokinetic Tables | 111 |
| | 13.11.10 | .Pharmacokinetic Figures | 112 |
| | 13.11.11 | .Biomarker Tables | 112 |
| | 13.11.12 | .Biomarker Figures | 115 |
| | 13.11.13 | .ICH Listings | 117 |
| | 13.11.14 | .Non-ICH Listings | 120 |
| 13.12. | Appendix | c 12: Example Mock Shells for Data Displays | 121 |

## 1. INTRODUCTION

The purpose of this reporting and analysis plan (RAP) is to describe the analyses to be included in the Clinical Study Report for Protocol 116027:

| Revision Chronology | Revision Chronology: | |
|---------------------|----------------------|--------------|
| 2012N154810_00 | 22-Aug-2013 | Original |
| 2012N154810_01 | 04-Oct-2013 | Amendment 01 |
| 2012N154810_02 | 14-Jan-2014 | Amendment 02 |
| 2012N154810_03 | 01-Apr-2014 | Amendment 03 |
| 2012N154810_04 | 31-Aug-2015 | Amendment 04 |
| 2012N154810_05 | 03-Dec-2015 | Amendment 05 |
| 2012N154810_06 | 12-Sep-2017 | Amendment 06 |

#### 2. KEY PROTOCOL INFORMATION

A total of approximately 71 subjects (10 in the treatment holiday group, 26 in the treatment control group, and 35 in the long-term discontinuation group) will be enrolled in this study. The total sample size is based on practical considerations on the availability of subjects from other ongoing belimumab studies, rather than on statistical considerations. Since this is a non-randomized study, results will be descriptive only, and not intended to be inferential. No power calculations were made in the determination of sample size for this study. However, the total of subjects is expected to provide adequate information to characterize time to SLE flare.

Table 1 Flare Rates from Pooled BLISS Studies

| ISE Table | Analysis | Placebo | 1 mg/kg | 10 mg/kg |
|---|---|---|---|---|
| T57 | Percentage of Subjects<br>with Flare Over 52<br>Weeks | 81.5% | 74.6% | 74.6% |
| TAC411 | Percentage of Subjects<br>with Flare Over 52<br>Weeks Post Week 24 | 68.5% | 54.7% | 57.5% |
| TAC613 | Percentage of Subjects<br>with Flare Over 52<br>Weeks Among SRI Wk<br>52 Responders | 73.4% | 69.8% | 67.4% |

## 2.1. Changes to the Protocol Defined Statistical Analysis Plan

Changes from the originally planned statistical analysis specified in the protocol are outlined in Table 2.

Table 2 Changes to Protocol Defined Analysis Plan

| Protocol F | | | Reporting & Analysis Plan | | |
|---|---|---|---|---|---|
| Statistical Analysis Plan | | Statistical Analysis Plan | | Rationale for Changes | |
| • | Partial prothrombin time (PTT) is collected | • | Activated partial prothrombin time (aPTT) time is analyzed | • | aPTT was collected instead of PTT |
| • | Section 8.1.3 states that for the primary analysis of the additional efficacy and biomarkers, the baseline will be defined as study Day 0 of the original parent study. Additionally, for some of the endpoints, a secondary analysis will be performed by defining the baseline as Day 0 of the BEL116027 study. | • | The baseline for each endpoint is defined per Section 6.1 of the protocol. | • | The protocol was inconsistent in the definition of baseline. See RAP Section 5.3 for clarification |
| • | Immunogenicity is listed as a secondary endpoint in Protocol Section 6.1.2., but as an exploratory laboratory parameter in the Time and Events table. | • | Immunogenicity is defined as a secondary endpoint. | • | The protocol was inconsistent, so the correct category was used in the RAP. |
| • | Renal flares are not listed as an endpoint in Protocol Section 6.1.2 nor described in Protocol Section 8, but are defined in Protocol Section 6.1.4 | • | Renal flares are included as an exploratory endpoint in RAP Section 2.2. | • | The protocol was inconsistent, so the endpoint was correctly specified in the RAP. |
| • | The definition of renal flare contained a typographical error and referenced an increase rather than a decrease in GFR. This was corrected in a note to file. | • | The RAP specifies the correct definition, referencing a decrease in GFR. | • | The protocol was incorrect. |
| • | Protocol Section 6.1.3 lists percent change in PGA. | • | The RAP specifies change from baseline in PGA instead. | • | Change from baseline is more clinically relevant and interpretable, particularly in the case of low baseline scores. |
| • | Protocol Section 6.1.2 lists one time interval for percent change in B-cell subsets from Week 24, i.e., Week 24 to 52. | • | In addition to this, the RAP specifies percent change from Week 24 to 32 and Week 24 to 40. | • | The additional time intervals facilitate interpretation of the changes following the treatment holiday phase. |
| • | The protocol Section 6.1.2 does not list the CD19+ B-cell subset. | • | The RAP adds the CD19+<br>B-cell subset. | • | This subset is collected and clinically important. |
| • | The protocol Section 6.1.3 Other Endpoints includes percent change in prednisone dose and percent of subjects with prednisone dose reduced to <7.5mg/day from ≥7.5mg/day | • | These two exploratory endpoints were not analysed | • | The two secondary prednisone endpoints (Protocol Section 6.1.2) will be analysed as they are most descriptive in that they assess daily prednisone use. Given the reduced sample size from |

| Protocol | Reporting & Analysis Plan | |
|---|---|---|
| Statistical Analysis Plan | Statistical Analysis Plan | Rationale for Changes |
| Section 6.1.2 lists percent change from baseline in B-Cells, immunoglobulins and autoantibodies | Change from baseline will also be presented for these parameters. | the original protocol, these two endpoints allow sufficient evaluation of the impact of the treatment holiday. Change from baseline added based on regulatory feedback on other studies in the belimumab development |
| | | program. |

## 2.2. Study Objective(s) and Endpoint(s)

| Objectives | Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| Characterize the efficacy of a 24-week withdrawal followed by a 28-week reintroduction of intravenous belimumab therapy compared with uninterrupted intravenous belimumab therapy for 52 weeks in subjects with low SLE disease activity receiving belimumab 10 mg/kg plus standard of care, as measured by time to first flare. | Time to any SLE Flare Index flare. |
| Secondary Objectives | Secondary Endpoints |
| Evaluate the rate of any flare. | <ul> <li>Rate of any SLE Flare Index flare per subject year.</li> <li>Time to first SLE Flare Index severe flare.</li> </ul> |
| Assess safety. | <ul> <li>Adverse events</li> <li>AESI</li> <li>Laboratory parameters</li> <li>Vital signs</li> </ul> |
| Assess SLE disease activity. | <ul> <li>Number of subjects in the treatment holiday and long-term discontinuation group with evidence of rebound (defined as a SELENA SLEDAI score during the first 24 weeks that exceeds the baseline SELENA SLEDAI score in the subjects' respective original parent study).</li> <li>SELENA SLEDAI scores change from baseline.</li> </ul> |
| Assess immunogenicity. | Response (Negative, Transient Positive, Persistent Positive) by Visit and Across All Visits |
| Assess markers of autoimmune response (e.g., immunoglobulins, complement.) | <ul> <li>Change and Percent change from baseline in IgG, IgM, IgA, anti-dsDNA, ANA, C3, and C4.</li> <li>Shifts from baseline in IgG, IgM, IgA, anti-dsDNA, ANA, C3 and C4.</li> <li>Change and Percent change in absolute B cell subsets</li> </ul> |

| Objectives | Endpoints |
|---|---|
| | (CD19+, CD20+, CD20+/27+ memory, CD20+/27- naïve, CD20+/69+ activated, CD20+/138+ plasmacytoid, CD19+/27BRIGHT/38BRIGHT SLE subset and CD20-/138+ plasma cells) at Weeks 0, 8, 16, 24, 32, 40 and 52 and from Weeks 24 to 52. |
| Assess changes in corticosteroid use. | <ul> <li>Number of days of daily prednisone dose ≥7.5 mg/day and/or increased by 25% from Day 0 of this study to Week 24, from Day 0 of this study to Week 52, and from Week 24 to Week 52.</li> <li>Number of days of daily prednisone dose ≤7.5 mg/day and/or decreased by 25% from Day 0 of this study to Week 24, from Day 0 of this study to Week 52, and from Week 24 to Week 52.</li> </ul> |
| Exploratory/Other | Exploratory/Other Endpoints |
| | <ul> <li>Time to first renal flare</li> <li>Time to first renal flare among subjects with baseline proteinuria &gt;0.5g/24hr equivalent</li> <li>Change from Baseline in PGA</li> <li>Change and percentage change from Baseline in BLyS Protein</li> <li>SLICC/SDI</li> <li>Change from Baseline</li> </ul> |

## 2.3. Study Design



| Overview of Study Design and Key Features | |
|---|---|
| | this long-term safety data to regulatory authorities in the initial BLA and other marketing authorization submissions). Additional interim analyses may be required to support subsequent safety updates to regulatory authorities. No interim analyses were conducted. |
| Sample Size | The total target sample size was 71 subjects and 80 were enrolled. The target sample size for subjects in the treatment holiday and control groups was 10 (12 enrolled) and 26 (29 enrolled) subjects respectively. A target sample size of 35 (39 enrolled) subjects in the long-term discontinuation group was anticipated. |

Note: Subjects from China participated in BEL113750 OL phase rather than in BEL114333, and were therefore eligible to enter BEL116027 from BEL113750 OL, per a China country-specific protocol amendment 01.

## 2.4. Statistical Hypotheses / Statistical Analyses

Since this is a non-randomized study, results will be descriptive only, and any comparisons are not intended to be inferential.

## 3. PLANNED ANALYSES

## 3.1. Interim Analyses

The protocol indicated that an interim analysis of the data in this trial may be performed to support a submission to regulatory authorities relating to marketing authorization (e.g., to summarize and submit this long-term safety data to regulatory authorities in the initial BLA and other marketing authorization submissions). Additional interim analyses may be required to support subsequent safety updates to regulatory authorities. No interim analyses were conducted.

The SRT performs in stream adjudication of subject-level safety data for Adverse Events of Special Interest (AESIs; serious and non-serious) in accordance with the GSK Standard Operating Procedures (SOPs) and the belimumab Program Safety Analysis Plan (PSAP). AESIs include malignancy; serious hypersensitivity and post-infusion systemic reactions; potential opportunistic infections; other infections of interest but not generally considered opportunistic i.e. Mycobacterium Tuberculosis and Herpes Zoster; suicide/self-injury; and fatalities.

AESIs are flagged in the clinical trial database, according to SRT adjudication. The SRT performs a periodic review of instream study data (at least every 6 months), reviewing the cumulative incidence of AEs, SAEs, and adjudicated AESIs. These periodic reviews of cumulative adverse event incidence are compared with previous SRT reviews and where appropriate, the pivotal SLE pooled data to assess for any new safety signals.

## 3.2. Final Analyses

The final planned primary analyses will be performed after the database cleaning activities have been completed and final database release and database freeze has been declared by Data Management:

database cleaning activities have been completed and final database release and database freeze has been declared by Data Management.

In this open-label, non-randomized study, for dispensing of study drug, randomisation codes have been distributed according to RandAll NG procedures.

## 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Screened | Comprises all subjects who enroll in the study, including screen failures | Study population |
| Intent-To-Treat | Comprises all subjects who enroll in the study, | Study population |
| | excluding screen failures. | Efficacy |
| | | Safety |
| | | Biomarker |
| PK | Comprises all subjects included in the ITT population for whom at least one post belimumab treatment PK sample was obtained and analyzed. | • PK |

#### 1. NOTES:

• Please refer to Appendix 11: List of Data Displays which details the population to be used for each display being generated.

#### 4.1. Protocol Deviations

Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be identified in the Protocol Deviation Management Plan (PDMP).

Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the PDMP.

- Data will be reviewed prior to freezing the database to ensure all important deviations are captured and categorised on the protocol deviations dataset.
- This dataset will be the basis for the summaries and listings of protocol deviations.

Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarised and listed

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

## 5.1. Study Treatment Descriptors

| Treatment Group Descriptions | | | |
|---|---|---|---|
| | RandAll NG | Data Displays for Report | ing |
| Group<br>Code | Group Description | Description | Order [1] |
| 3 | Long Term Discontinuation Group | Long-term Discontinuation | 1 |
| 2 | Control Group | Treatment Control | 2 |
| 1 | Treatment Holiday Group | Treatment Holiday | 3 |

#### NOTES:

- Order represents treatments being presented in TFL, as appropriate. Some Tables will only present TC and TH groups.
- 2. In applicable data listings, Screen Failures will be presented first followed by LTD, TC and TH.

#### 5.2. Parent Studies

Subjects were eligible to enter BEL116027 from one of four continuation studies, having entered the continuation study from a respective parent study. The possible study participation sequences are as follows:

| Parent Study | <b>Continuation Study</b> | Subjects |
|---|---|---|
| BEL113750 DB <sup>1</sup> | BEL113750 OL1 | Subjects from China |
| BEL112341 <sup>2</sup> | BEL114333 | Some subjects from Japan |
| BEL113750 | BEL114333 | Subjects from Korea and some subjects from Japan |
| BEL110751 | BEL112233 (C1066) | Subjects from US |
| LBSL02 | LBSL99 (BEL112626) | Subjects from US |

- 1. BEL113750 was both the parent and continuation study number for subjects enrolled in China.
- 2. Subjects from Japan who participated in study BEL112341 were eligible to enrol into the BEL114333 continuation phase per a BEL114333 protocol amendment, to allow them continued access to study agent until belimumab was commercially available in Japan.

#### 5.3. Baseline Definitions

#### 5.3.1. Baseline Definitions<sup>1</sup>

The baseline (BL) definition is dependent upon the endpoint being analyzed.

• For the SELENA SLEDAI (including rebound), immunoglobulins, autoantibodies, complement, BLyS and B-cell endpoints, baseline is defined as the Day 0 assessment in the subject's respective parent study, prior to exposure with study treatment (whether placebo or belimumab). Baseline data for these

- parameters will be extracted from the ADaM data sets from the double blind study (LBSL02, BEL110751, BEL113750 or BEL112341) from which the patients are enrolled.
- For the SLE flares, SLE severe flares, SLICC, prednisone (7 day average prior to Day 0), PGA, and immunogenicity<sup>2</sup>, endpoints, baseline is the Day 0 assessment in BEL116027.
- For other endpoints, baseline is the Day 0 assessment in BEL116027<sup>2</sup>.

<sup>1</sup>Feeder study BEL114333 database had not yet completed at the time of BEL116027 Last Patient Last Visit. Consequently, baseline data for BEL114333 patients has not been fully cleaned when extracted from that study's database for reporting.

<sup>2</sup>Assessments covered for both Day 0 in BEL116027 and the Exit/Follow-up visit of the feeder continuation studies were only to be performed once and were to be recorded in the appropriate case report forms for each study. For Day 0 values not recorded in BEL116027 CRF but exist in the feeder study, the data will be extracted from the appropriate feeder study for inclusion in analysis

In the displays, the baseline value/visit will be denoted as Baseline.

See Section 13.4.1 for a diagram depicting the baseline definitions and phases.

## 5.3.2. Derivations and Handling of Missing Baseline Data

| Definition | Reporting Details |
|---|---|
| Change from Baseline | = Post-Dose Visit Value – Baseline |
| % Change from Baseline | = 100 x [(Post-Dose Visit Value – Baseline) / Baseline] |
| Maximum Change from Baseline | = Calculate the change from baseline at each given timepoint |
| | and determine the maximum change |

#### NOTES:

- Unless otherwise specified, the baseline definitions specified in Section 5.3.1 Baseline Definitions will be used for derivations for endpoints / parameters and indicated on summaries and listings.
- Unless otherwise stated, if baseline data is missing no derivation will be performed and baseline will be set to missing.

#### 5.4. Multicentre Studies

In this multicentre global study, enrolment will be presented by investigative site, and in selected displays by country and investigative site.

Since this is a non-randomized study, results will be descriptive only, and there will be no methods applied to address multiple centers.

# 5.5. Other Considerations for Data Analyses and Data Handling Conventions

Other considerations for data analyses and data handling conventions are outlined in the appendices:

| Section | Component |
|---|---|
| 13.1 | Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population |
| 13.2 | Appendix 2: Schedule of Activities |
| 13.3 | Appendix 3: Assessment Windows |
| 13.4 | Appendix 4: Study Phases and Treatment Emergent Adverse Events |
| 13.5 | Appendix 5: Data Display Standards & Handling Conventions |
| 13.6 | Appendix 6: Derived and Transformed Data |
| 13.7 | Appendix 7: Reporting Standards for Missing Data |
| 13.8 | Appendix 8: Values of Potential Clinical Importance |
| 13.9 | Appendix 9: Adverse Events of Special Interest |
| 13.11 | Appendix 10: Abbreviations & Trade Marks |
| 13.12 | Appendix 11: List of Data Displays |
| 13.12 | Appendix 12: Example Mock Shells for Data Displays |

#### 6. STUDY POPULATION ANALYSES

# 6.1. Overview of Planned Demography, Baseline Characteristics and Medical History Analyses

The study population analyses including analyses of subject's disposition, protocol deviations, demographic and baseline characteristics, medical conditions, prior and concomitant medications, and exposure and treatment compliance will be based on the ITT population, or for the Screened population where specified. Data will be presented by treatment group and for all subjects combined, unless otherwise specified.

Full details of data displays being presented in Appendix 11: List of Data Displays.

Completion and withdrawal status by treatment phase is defined in Section 13.6.2.

## 6.2. Baseline Disease Activity and Other Baseline Endpoints

A summary of baseline disease activity will be provided, including counts and percentages for categorical endpoints and descriptive statistics for the continuous endpoints and scores.

Table 3 provides indicators of baseline disease activity that will be summarized. Some of these parameters will be summarized on the by visit summary for that parameter according to the table specifications.

Table 3 Baseline Disease Activity Endpoints

| Endpoint | Categories & Summaries at Baseline |
|---|---|
| SELENA-SLEDAI category | Continuous |
| | Categorical |
| | • 0, 1, 2, 3 |
| SELENA SLEDAI by organ domain | Categorical |
| and item at baseline | Presented if Yes |
| Complement & BLyS Levels | Complement C3 and C4 (mg/dL) |
| | Continuous |
| | Categorical |
| | Positive, Negative |
| | Low, Normal, High |
| | (See Section 13.6.6 for definitions) |
| | BLyS Protein [ng/mL] |
| | Continuous |
| | Categorical |
| | Below LLOQ: <0.061 ng/mL for China samples and <0.02048 ng/mL for all others |
| SLE Flare Index | Categorical |
| | At least 1 flare, At least 1 severe flare |
| PGA | Continuous |
| | Categorical |
| | • 0-1, >1 – 2.5, > 2.5 |
| SLICC/ACR Damage Index | Continuous |
| | Categorical |
| | • 0, 1, > 1 |

| Endpoint | Categories & Summaries at Baseline |
|---|---|
| Proteinuria (based on spot urine using | Continuous |
| protein: creatinine mg/mg ratio) | Categorical (units are g/24hr equivalent) |
| | • ≤ 0.5, > 0.5 |
| | • Subcategories of > 0.5 |
| | <ul><li>&gt;0.5 - &lt; 1</li></ul> |
| | • 1-<2 |
| | • ≥2 |
| B cells: | Continuous |
| CD19+ | |
| CD20+ | |
| CD20+/27+ memory | |
| CD20+/27- naïve | |
| CD20+/69+ activated | |
| CD20+/138+ plasmacytoid<br>CD19+/27 <sup>BRIGHT</sup> /38 <sup>BRIGHT</sup> SLE subset | |
| CD20-/138+ plasma | |
| CD20-/130+ piasina | |
| Autoantibody Levels | Anti-dsDNA [IU/mL] |
| · | Continuous |
| | Categorical |
| | Positive: >=30 IU/mL |
| | Negative: <30 IU/mL |
| | ANA [Titer] |
| | Continuous |
| | Categorical |
| | Positive: Index >=0.80 |
| | Negative: Index < 0.80 |
| | aCL Status |
| | Categorical |
| | Positive, Negative, Missing (See Section 13.6.6 for |
| | definitions) |
| anti-dsDNA and/or ANA positive | Categorical |
| | Yes, No |
| Immunoglobulin Levels (IgG, IgA, and | Continuous |
| IgM [g/L]) | Categorical |
| | <u>lgG</u> |
| | • Low: < 6.94 g/L, High: > 16.18 g/L |
| | <u>lgM</u> |
| | Low: < 0.48 g/L, High: > 2.71 g/L |
| | <u>lgA</u> |
| | • Low: < 0.81 g/L, High: > 4.63 g/L |

| Endpoint | Categories & Summaries at Baseline |
|---|---|
| Allowable SLE Medication Usage | Categorical: Steroid Only Immunosuppressant Only Anti-malarial Only Steroid and Immunosuppressant Only Steroid and Anti-Malarial Only Immunosuppressant and Anti-Malarial Only Steroid and Immunosuppressant and Anti-malarial Traditional Chinese Medicine - Glycosides of Paeony/Tripterygium |
| Average daily prednisone dose (mg/day) at baseline | Continuous Categorical • 0, >0 to ≤7.5, >7.5 |
| PT/aPTT | Continuous |

# 6.3. Study Population Data for Maintenance Phase Subject Profile

Basic demography information will be listed on the subject profile.

## 7. EFFICACY ANALYSES

For all efficacy analyses, results for the TH group will be presented for the treatment holiday (TH) and re-start (RS) phases separately.

## 7.1. Primary Efficacy Analyses

## 7.1.1. Endpoint / Variables

The time to the first SFI flare over 52 weeks will be estimated for the treatment groups using the product-limit method.

Analyses of SFI flare (defined as mild, moderate, or severe) will be performed on the SELENA SLEDAI SLE flare index. Note: Flares in this study are analysed using the modified SLE flare index where severe flares that are triggered only by an increase in SELENA SLEDAI score to greater than 12 are not categorized as severe in the analysis.

## 7.1.2. Summary Measure

Only post-baseline flares will be considered in these analyses. Flares (not subjects) occurring on the Day 0 visit date should be removed from the analysis set prior to determining the first flare.

Data observed at or prior to the baseline visit (see Section 5.3.1) will not be included in this analysis.

Time to first SFI flare is defined as the number of days from baseline date (see Section 5.3.1) to the date the subject has a flare (event date – baseline visit date + 1).

See Section. 13.6.3 for additional details.

## 7.1.3. Population of Interest

The primary efficacy analyses will be based on ITT population.

## 7.1.4. Strategy for Intercurrent (Post-Randomization) Events

The disposition of subjects as it relates to intercurrent events is defined as follows:

| | Event | |
|---|---|---|
| Subject Disposition | Met | Event Date [2] |
| Subject has a SFI flare or takes a prohibited medication | | |
| Subject has a SFI flare during the study | Yes | Date of first SFI flare |
| [1] | | |
| Subject takes a prohibited medication [1] | Yes | Date of prohibited medication |
| Subject does not have a SFI flare and did not take a prohibited medication. | | |
| Subject withdraws from the study or is | No | Censored at last available date where |
| lost to follow-up | | flare is assessed. |
| Subject dies during the study | No | Censored at date of death. |

| Subject completes the study | No | Censored at last study visit where flare is |
|---|---|---|
| | | assessed. |

<sup>[1]</sup> If a subject has a SFI flare and takes a prohibited medication, the event date is the earliest of the first SFI flare date and takes a prohibited medication date.

## 7.1.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 11: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 7.1.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

The table will display the number and percentage of subjects with a SFI flare, as well as the median, 25th, and 75th percentile of days to first SFI flare, estimated using the product-limit method. For subjects who experience a SFI flare, the study day of the SFI flare will be summarized and the table will display the median, 25th and 75th percentiles and minimum and maximum.

A cumulative incidence curve for time to first SFI flare will also be produced for the 52-week treatment phase.

## 7.2. Secondary Efficacy Analyses

## 7.2.1. Endpoint / Variables

#### 7.2.1.1. Rate of Flares

The unadjusted rate of flares per subject-year over 52 weeks will be summarized by treatment group.

#### 7.2.1.2. First Severe SFI Flare

The time to the first severe SFI flare over 52 weeks will be estimated for the treatment groups using the product-limit method.

#### 7.2.1.3. Rebound

Rebound is defined as a SELENA SLEDAI score during the first 24 weeks that exceeds the baseline SELENA SLEDAI score in the subject's respective original parent study.

#### 7.2.1.4. SELENA SLEDAI Scores

SELENA SLEDAI assessments consist of 24 individual weighted items in which signs and symptoms, laboratory tests, and physician's assessment for each of 8 organ systems are given a weighted score and summed if present (marked 'Yes') at the time of the visit or in the preceding 10 days. The maximum theoretical score is 105 (all 24 descriptors

<sup>[2]</sup> If a subject meets multiple criteria, then the event date is the earliest date.

present simultaneously) with 0 indicating inactive disease (marked 'No'), but in practice few subjects have scores > 45 [Buyon, 2005; Petri, 2005].

See Section 13.6.3 for further details.

#### 7.2.2. Summary Measure

#### 7.2.2.1. Rate of Flares

The total number of flares, total subject-years of follow-up in the time interval, and the unadjusted rate per subject-year will be presented.

#### 7.2.2.2. First Severe SFI Flare

See Section 7.1.2.

#### 7.2.2.3. Rebound

The frequencies and percentages of subjects who rebound will be presented by visit through the Week 24 visit, and at any time during the first 24 weeks.

#### 7.2.2.4. SELENA SLEDAI Scores

Summary statistics for the change from baseline in SELENA SLEDAI scores will be presented at each visit in the 52-week treatment phase.

#### 7.2.2.5. Changes in Corticosteroid Use

The frequencies and percentages of subjects who meet each definition will be presented at each visit in the 52-week treatment phase. Steroid doses will be converted to the prednisone-equivalent dose per the derivations in Section. 13.6.3

#### 7.2.3. Population of Interest

The secondary efficacy analyses for all endpoints will be based on the ITT population.

For rebound, the analysis also will be performed by the SELENA SLEDAI score at the BEL116027 Day 0 visit, categorized as  $\leq 3$  and  $\geq 3$ .

## 7.2.4. Strategy for Intercurrent (Post-Randomization) Events

#### 7.2.4.1. Rate of Flares and First Severe SFI Flare

See Section 7.1.4.

If a subject withdraws from the study, dies or takes a prohibited medication, the subject will be considered as having a SFI flare.

#### 7.2.4.2. Rebound and SELENA SLEDAI Scores

Missing data will be imputed using the principle of Last Observation Carried Forward (LOCF). For the TH group, LOCF will not be applied across the TH and RS phases. If an individual SS item data is missing at the first timepoint in the RS phase, the item will be considered not present.

## 7.2.4.3. Changes in Corticosteroid Use

# 7.2.4.3.1. Number of days of daily prednisone dose ≥7.5 mg/day and/or increased by 25%

The Dropout (DO)/Prohibited Medication (PM)=Non-responder (NR) imputation will be applied. If a subject withdraws from the study and/or receives a protocol-prohibited medication, the subject will be considered to have met this endpoint criteria (i.e, dose ≥ 7.5 mg/day and/or increased by 25%) after the date of dropout or the date that the medication is started, whichever comes first, up until the visit date, and for those days in intervals for subsequent attended visits. Before this date, the evaluated endpoint will be assessed using available data.

## 7.2.4.3.2. Number of days of daily prednisone dose ≤7.5 mg/day and/or decreased by 25%

The Dropout (DO)/Prohibited Medication (PM)=Non-responder (NR) imputation will be applied. If a subject withdraws from the study and/or receives a protocol-prohibited medication, the subject will be considered a non-responder for this endpoint criteria (i.e., dose >7.5 mg/day and/or did not decreased by 25%) after the date of dropout or the date that the medication is started, whichever comes first, and for those days in intervals for subsequent attended visits. Before this date, the evaluated endpoint will be assessed using available data.

## 7.2.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 11: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 7.2.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

## 7.3. Exploratory Efficacy Analyses

## 7.3.1. Endpoint / Variables

## 7.3.1.1. Physician Global Assessment (PGA)

The change from baseline in PGA score will be assessed at each visit in the 52-week treatment phase. See Section. 13.6.3 for additional details on the instrument.

#### 7.3.1.2. SLICC/SDI

The change from baseline in SLICC/SDI score will be assessed at each visit in the 52-week treatment phase.

#### 7.3.1.3. Renal Flare

The time to the first renal flare over 52 weeks will be estimated for the treatment groups using the product-limit method. See Section 13.6.3 for additional details.

## 7.3.2. Summary Measure

#### 7.3.2.1. Physician Global Assessment (PGA) and SLICC/SDI

These endpoints will be analyzed using summary statistics.

#### 7.3.2.2. Renal Flares

Only post-baseline renal flares will be considered in these analyses. Renal flares (not subjects) occurring on the Day 0 visit date should be removed from the analysis set prior to determining the first renal flare.

Data observed at or prior to the baseline visit (see Section 5.3.1) will not be included in this analysis.

Time to first renal flare is defined as the number of days from baseline date (see Section 5.3.1) to the date the subject has a renal flare (event date – baseline visit date + 1).

## 7.3.3. Population of Interest

The analyses for all exploratory endpoints will be based on the ITT population.

For renal flares, the analysis will be repeated for subjects with baseline proteinuria proteinuria >0.5g/24hr equivalent.

## 7.3.4. Strategy for Intercurrent (Post-Randomization) Events

#### 7.3.4.1. Physician Global Assessment (PGA)

Missing data will be imputed using LOCF. For the TH group, LOCF will not be applied across the TH and RS phases.

#### 7.3.4.2. SLICC/SDI

Missing data due to study withdrawal will be imputed using LOCF. For the TH group, LOCF will not be applied across the TH and RS phases.

The SLICC/ACR Damage Index increases over time. Once a subject meets the criteria for positive scoring of an item, that item should always be marked as present, even if the subject subsequently recovered.

In the event the SLICC/ACR Damage Index is scored inconsistently (a decrease relative to previous items has occurred) and the data are unable to be queried and/or corrected, a worst observation carried forward (WOCF) approach will be used at the item level for the SLICC/ACR Damage Index questions. These WOCF values will then be used to calculate the total score which will be the value summarized and displayed for reporting.

#### 7.3.4.3. Renal Flare

The disposition of subjects as it relates to intercurrent events is defined as follows:

| Subject Disposition | Event Met | Event Date [2] |
|---|---|---|
| Subject has a renal flare or takes a prohibited medication | | |
| Subject has a renal flare [1] | Yes | Date of first renal flare |
| Subject takes a prohibited | Yes | Date of prohibited medication |
| medication [1] | | |
| Subject does not have a renal flare and did not take a prohibited medication | | |
| Subject withdraws | No | Censored at last flare |
| | | assessment date |
| Subject dies | No | Censored at date of death |
| Subject completes | No | Censored at the Week 52 |
| | | study visit |

<sup>[1]</sup> If a subject has a renal flare and takes a prohibited medication, the event date is the earliest of the first renal flare date and takes a prohibited medication date.

## 7.3.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 11: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 7.3.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

## 7.4. Efficacy Data for Maintenance Phase Subject Profile

Flare data will be listed on the subject profile.

<sup>[2]</sup> If a subject meets multiple criteria, then the event date is the earliest date.

## 8. SAFETY ANALYSES

The safety analyses will be based on the ITT population, unless otherwise specified.

## 8.1. Adverse Events Analyses

Adverse events analyses including the analysis of adverse events (AEs), serious adverse events (SAEs), and other significant AEs will be based on GSK Core Data Standards. The details of the planned displays are provided in Appendix 11: List of Data Displays.

Adverse events will be coded to the current MedDRA dictionary version available at the time of reporting.

Only treatment emergent AEs will be summarized (see Section 13.4.1). Any AEs that were ongoing in the upon entry into this will be listed and flagged with a footnote

An overall summary of AEs will be presented showing the number (%) of subjects with at least one of the following: AE, related AE, SAE, severe AE, SAE and/or severe AE, AE resulting in study treatment discontinuation, and deaths.

The number of events and the number (%) of subjects experiencing an AE by SOC, SOC and PT, and PT will be summarized for each of the AE categories below.

- A11
- Serious
- Severe
- Study agent Related
- Resulting in discontinuation of study treatment

The data will be sorted by overall decreasing frequency of the SOC, by overall decreasing frequency of the SOC and then decreasing frequency of PT within the SOC, and by overall decreasing frequency of the PT, as applicable. Only SOCs with observed AE PTs will be presented. If the frequency for any two or more adverse events is equal, the events will be presented in alphabetical order by SOC/PT as applicable.

Summaries of AEs frequency by SOC and severity will also be provided. For these displays, the number and percentage of subjects will be summarized as mild, moderate, or severe based on the maximum severity observed across all PTs within the SOC for a given subject.

The hierarchical relationship between MedDRA SOCs, PTs, and verbatim text will be displayed in a table for all AEs.

A listing of which subjects reported each AE will be produced. AEs will be grouped and sorted by SOC and PT. A listing of Infusion Related Systemic Reactions will be produced.

## 8.2. Adverse Events of Special Interest Analyses

## 8.2.1. Endpoint / Variables

## 8.2.1.1. Adverse Events of Special Interest

A comprehensive list of MedDRA terms based on clinical review will be used to identify each type of event. Changes to the MedDRA dictionary may occur between the start of the study and the time of reporting and/or emerging data from on-going studies may highlight additional adverse events of special interest, therefore the list of terms to be used for each event of interest and the specific events of interest will be based on the safety review team (SRT) agreements in place at the time of reporting. The details of the planned displays are provided in Appendix 11: List of Data Displays.

Adverse events of special interest for belimumab have been identified over the course of the development program. The Benlysta Program Safety Analysis Plan (PSAP) includes the definitions and adjudication criteria for the AESI. The definitions are based on standard and custom MedDRA queries (SMQs and CMQs). Categorizations for the AESI are listed in Section 13.9.

GSK will adjudicate neoplasms of unspecified malignancy, opportunistic infections, herpes zoster, serious suicide, and serious PISR events as described in the PSAP. In addition, GSK will review malignancy events to prevent counting an event multiple times in the case where a given malignancy has multiple events (e.g., a diagnostic test and the diagnosis). GSK will review all fatal events and assign a category of death.

#### 8.2.1.2. Post-infusion systemic reactions by infusion

For the TH group in the RS phase, summaries of post-infusion systemic reactions will be presented by the first six infusions in the RS phase and PT for the following categories:

- Post-Infusion Systemic Reactions per Anaphylactic Reaction CMQ broad search (on the day of the infusion or within 3 days after the infusion)
- Serious Post-Infusion Systemic Reactions per Anaphylactic Reaction CMQ broad search (on the day of the infusion or within 3 days after the infusion)
- Serious Acute Post-Infusion Systemic Reactions/Hypersensitivity per GSK adjudication
- Serious Delayed Acute Hypersensitivity Reactions per GSK adjudication
- Serious Delayed Non-Acute Hypersensitivity Reactions per GSK adjudication

## 8.2.2. Summary Measure

#### 8.2.2.1. Adverse Events of Special Interest

An overall summary of AESIs by category will be presented, and each specific category of AESI will be presented separately by PT. The number and percentage of subjects with at least one occurrence and the number of events will be presented.

Infection AESIs that are serious, severe, serious/severe, and that lead to discontinuation will be presented by category and PT.

#### 8.2.2.2. Post-infusion systemic reactions by infusion

The number and percentage of subjects with at least one occurrence and the number of events will be presented.

#### 8.2.3. Population of Interest

The analyses will be based on the ITT population.

#### 8.2.4. Strategy for Intercurrent (Post-Randomization) Events

For both endpoints, observed data will be used with no imputation.

#### 8.2.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 11: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 8.2.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

## 8.3. Clinical Laboratory Analyses

Laboratory evaluations including the analyses of chemistry laboratory tests, hematology laboratory tests, urinalysis, and liver function tests will be based on GSK Core Data Standards. The details of the planned displays are in Appendix 11: List of Data Displays.

An issue was identified at Q2 Solutions (central lab) in Valencia, California, USA, regarding equipment malfunction which affected some serum creatinine results reported from one of the analyzers used at the lab. Unusually high serum creatinine results were noted for two different GSK clinical trials, and further investigation revealed one of the analyzers had been producing intermittent high serum creatinine results between 01 October 2016 to 13 January 2017, potentially due to an intermittent wash line blockage of the analyzer. BEL116027 investigators were notified of this issue by a Dear Investigator Letter (DIL) 22 February 2017. The subsequent evaluation concluded that there was no impact on data integrity and patient safety for clinical trial BEL116027. Therefore, there will be no modification to the analysis of serum creatinine. BEL116027 investigators were notified by a follow up DIL dated 25 July 2017, and the root cause was identified as a sporadic failure of the wash system due to debris causing intermittent obstruction.

Baseline is defined as described in Section 5.2.

A list of laboratory parameters collected and definition of the toxicity grades are provided in Appendix 8: Values of Potential Clinical Importance.

Listings will be generated for all laboratory results, and additionally for Grade 3 or Grade 4 laboratory toxicity results.

Line graphs will be produced for each analyte displaying the mean value by visit and treatment group.

## 8.3.1. Endpoint / Variables

## 8.3.1.1. Clinical Laboratory Results

Laboratory parameters which are continuous numeric values will be analyzed using summary statistics, and those with categorical results will be summarized using frequencies and percentages.

## 8.3.1.2. Clinical Laboratory Toxicity Grades

The endpoints evaluated will be:

- Worst toxicity grade
- Worsening by at least 2 toxicity grades

Toxicities will be reported as derived by the central laboratory, as protocol toxicity grading was applied.

For potassium, glucose, calcium, and sodium, toxicities are bi-directional (i.e., high and low directions) and both will be summarized by name of the toxicity.

- Potassium: hypokalemia, hyperkalemia
- Glucose: hypoglycemia, hyperglycemia
- Calcium: hypocalcemia, hypercalcemia
- Sodium: hyponatremia, hypernatremia

For example, calcium will have two toxicity sections, one for hypocalcemia and one for hypercalcemia and mapped to their high or low form as:

- RESULT < (LLN+ULN)/2 = "Hypo" toxicity
- RESULT > (LLN+ULN)/2 = "Hyper" toxicity

#### 8.3.1.3. Clinical Laboratory Reference Range Shifts

For laboratory tests without toxicity grades, shifts relative to the normal range will be summarized for each analyte as shifts 'to low' and shifts 'to high.'

For the 'to low category' the percentage of subjects with at least one low post-baseline value relative to the baseline (i.e. baseline and post baseline data available) will be displayed using the categories: no shift to low and normal/high to low.

For the 'to high category' the percentage of subjects with at least one high post-baseline value relative to baseline (i.e. baseline and post baseline data available) will be displayed using the categories: no shift to high and normal/low to high.

A laboratory value that is above the testing laboratory's normal range will be considered a high abnormal laboratory value. A laboratory value that is below the testing laboratory's normal range will be considered a low abnormal value.

#### 8.3.1.4. Immunoglobulin Results Relative to the Lower Limit of Normal

Immunoglobulins (IgG, IgA, IgM) will be classified relative to the reference range for the following categories: < LLN and  $\ge$  LLN.

## 8.3.2. Summary Measure

## 8.3.2.1. Clinical Laboratory Results

Laboratory parameters which are continuous numeric values will be analyzed using summary statistics, and those with categorical results will be summarized using frequencies and percentages. Results will be presented by visit during the 52-week treatment phase, and at any time post-baseline where specified.

#### 8.3.2.2. Clinical Laboratory Toxicity Grades

The frequencies and percentages of subjects meeting each of the toxicity grade endpoints will be summarized by visit during the 52-week treatment phase, and at any time post-baseline where specified.

#### 8.3.2.3. Clinical Laboratory Reference Range Shifts

The frequencies and percentages of subjects meeting each shift criteria will be summarized by visit during the 52-week treatment phase.

## 8.3.2.4. Immunoglobulin Results Relative to the Lower Limit of Normal

The frequencies and percentages of subjects who are <LLN and ≥LLN will be summarized by visit during the 52-week treatment phase. The analyses will be repeated for the subgroup of patients who are ≥LLN and who are <LLN at baseline, respectively.

#### 8.3.3. Population of Interest

For all clinical laboratory endpoints, the analyses will be based on the ITT population.

## 8.3.4. Strategy for Intercurrent (Post-Randomization) Events

For all clinical laboratory endpoints, observed data will be used with no imputation.

#### 8.3.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 11: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 8.3.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

## 8.4. Other Safety Analyses

The analyses of non-laboratory safety test results including immunogenicity and vital signs will be based on GSK Core Data Standards, unless otherwise specified. The details of the planned displays are presented in Appendix 11: List of Data Displays.

#### 8.4.1. Endpoint / Variables

#### 8.4.1.1. Immunogenicity

Serum samples for anti-belimumab antibody measurements will be obtained from subjects per the protocol

For the immunogenicity assessment, two types of antibody assays will be performed, i.e. a binding assay and neutralizing assay. For the binding assay, there will be 3-testing steps. A screening assessment is performed which produces a result of positive or negative. For samples with a positive screening result, a confirmation assay is then carried out, which also produces a result of positive or negative. For samples with a positive confirmation result, a titer value will also be obtained to quantify the degree of binding in a titration assay step. Patients will be viewed as positive for the binding assay if the confirmation assay was positive. Subjects, who tested positive for the binding assay, will be tested for the neutralizing assay, which again produces a result of positive or negative.
#### 8.4.1.2. Vital signs

Vital signs will be collected per the protocol. Parameters along with units for reporting are listed below

| Vital Sign Parameter<br>(Units) |
|-------------------------------------------|
| Systolic Blood Pressure (sitting) (mmHg) |
| Diastolic Blood Pressure (sitting) (mmHg) |
| Heart Rate (beats/min) |
| Temperature (C) |
| Weight (kg) |
| BMI (kg / m <sup>2</sup> ) |

## 8.4.2. Summary Measure

## 8.4.2.1. Immunogenicity

Immunogenic response will be summarized by visit and anytime postbaseline for the 52-week treatment phase.

Categories of response are Negative, Transient Positive (defined as a single positive response that does not occur at the final assessment, or Persistent Positive (defined as a positive response that occurs on at least 2 consecutive assessments or a single result at the final assessment).

#### 8.4.2.2. Vital signs

Change from baseline in vital signs will be presented using summary statistics by visit.

Baseline body mass index (BMI) will be calculated from weight and height measurements.

BMI 
$$(kg/m^2) = \frac{Weight (kg)}{[Height (m)]^2}$$

BMI will be derived at each visit using the baseline value for height and the weight at the visit. Since height is collected in centimeters (cm), it will be converted to meters (m) by dividing by 100 before using it in the formula above.

## 8.4.3. Population of Interest

For immunogenicity and vital signs endpoints, the analyses will be based on the ITT population.

## 8.4.4. Strategy for Intercurrent (Post-Randomization) Events

#### 8.4.4.1. Immunogenicity

Observed data will be used with no imputation.

## 8.4.4.2. Vital signs

Observed data will be used with no imputation. If weight or height is missing, then BMI will be missing.

## 8.4.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 11: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 8.4.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

## 8.5. Safety Data for Maintenance Phase Subject Profile

AE data, grade 3 or 4 laboratory data, and immunogenicity data will be listed on the subject profile.

## 9. PHARMACOKINETIC ANALYSES

## 9.1. Primary Pharmacokinetic Analyses

The primary PK analysis will be of the serum belimumab concentrations.

## 9.1.1. Endpoint / Variables

Refer Section 13.5.3 Reporting Standards for Pharmacokinetic.

## 9.1.2. Summary Measure

Descriptive statistics for serum belimumab concentrations will be displayed for each visit. The tables will display the mean value, standard deviation, 95% CI of mean, geometric mean, % CV, 95% CI of geometric mean, median, 25<sup>th</sup> and 75<sup>th</sup> percentiles, minimum and maximum.

## 9.1.3. Population of Interest

The primary pharmacokinetic analyses will be based on the PK population, unless otherwise specified.

## 9.1.4. Strategy for Intercurrent (Post-Randomization) Events

Observed data will be used with no imputation.

## 9.1.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 11: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 9.1.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

# 10. POPULATION PHARMACOKINETIC (POPPK) ANALYSES

Population Pharmacokinetic Analysis are not applicable to this study.

## 11. BIOMARKER ANALYSES

## 11.1. Primary Biomarker Analyses

## 11.1.1. Endpoint / Variables

Autoantibodies (anti-dsDNA, ANA), BLyS protein, B-cells (CD19+, CD20+, CD20+/27+ memory, CD20+/27-naïve, CD20+/69+activated, CD20+/138+plasmacytoid, CD19+/27BRIGHT/38BRIGHT SLE subset and CD20-/138+ plasma cells), immunoglobulins (IgG, IgA, and IgM), and complement (C3 and C4) will be assessed. See Section 13.6.6.2 for additional details.

## 11.1.2. Summary Measure

#### 11.1.2.1. B-Cells

For the B-cells, the change and percent change from baseline in the original parent study will be summarized at Weeks 0, 8, 16, 24, 32, 40 and 52 and from Week 24 to 32, Week 24 to 40, and Week 24 to 52.

## 11.1.2.2. Autoantibodies, Immunoglobulins and Complement

For autoantibodies, immunoglobulins and complement, the change and percent change from baseline in the original parent study to each visit including the Day 0 visit in the 52-week treatment phase will be assessed.

Shifts from baseline in IgG, IgM, IgA, anti-dsDNA, ANA, C3 and C4.

#### 11.1.2.3. BLyS Protein

The change and percent change from baseline in the original parent study to each visit in the 52-week treatment phase will be assessed.

## 11.1.3. Population of Interest

For all endpoints in Section 11.1.1, the primary biomarker analyses will be based on the ITT population.

## 11.1.4. Strategy for Intercurrent (Post-Randomization) Events

For all endpoints in Section 11.1.1, observed data will be used with no imputation.

## 11.1.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 11: List of Data Displays and will be based on GSK Data Standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 11.1.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

## 11.2. Biomarker Data for Maintenance Phase Subjects

By subject line plots for subjects who enter the maintenance phase for all visits for each B-cell parameter will be presented.

## 12. REFERENCES

Alarcón-Segovia D, Tumlin JA, Furie RA, et al for the LJP 394 Investigator Consortium. LJP 394 for the prevention of renal flare in patients with systemic lupus erythematosus. Arthritis Rheum. 2003;48(2):442–54.

Buyon JP, Petri MA, Kim MY, et al. The effect of combined estrogen and progesterone hormone replacement therapy on disease activity in systemic lupus erythematosus: A randomized trial. Ann Intern Med 2005;142(12 Pt 1):953-62.

Cockcroft DW, Gault MH. Prediction of creatinine clearance from serum creatinine. Nephron 1976;16:31-41.

Eibl MM, Rosen FS. Intravenous gamma globulin and plasmapheresis. In: Frank MM,editor. Samter's Immunologic Diseases (5th ed.). Boston:Little, Brown, 1995:1529-36.

Goldfarb NS, Avery RK, Goormastic M, Mehta AC, Schilz R, Smedira N, Pien L, HaugMT, Gordon SM, Hague LK, Dresing JM, Evans-Walker T, Maurer JR. Hypogammaglobulinemia in lung transplat recipients. Transplantation. 2001;71(2):242-6.

Petri M, Kim MY, Kalunian KC, et al. Combined oral contraceptives in women with systemic lupus erythematosus. N Engl J Med 2005;353(24):2550-8.

Yamini MH, Avery RK, Mawhorter SD, Young JB, Ratliff NB, Hobbs RE, McCarthyPM, Smedira NG, Goormastic M, Pelegrin D, Starling RC. Hypogammaglobulinemiafollowing cardiac transplantation: a link between rejection and infection. J Heart Lung Transplant. 2001;20(4):425-30.

## 13. APPENDICES

# 13.1. Appendix 1: Protocol Deviation

See Section 4.1 for details.

# 13.2. Appendix 2: Schedule of Activities

## 13.2.1. Protocol Defined Schedule of Events

## 13.2.2. Time and Events Table (Year 1)

| | Screen | | | | | | Tı | eatmen | t Holida | y Study | 1 | | | | | Follo | w-up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | | |
| Study Day | Up to -30 <sup>1</sup> | 0 2 | 28<br>±7d | 56<br>±7d | 84<br>±7d | 112<br>±7d | 140±<br>7d | 168<br>±7d | 196±<br>7d | 224<br>±7d | 252<br>±7d | 280±<br>7d | 308<br>±7d | 336<br>±7d | 364 ±7d or<br>Exit | 16-wk<br>±7d <sup>3</sup> | 6 mo<br>±7d |
| Study Week | | 0 | 4 | 8 | 12 | 16 | 20 | 24 | 28 | 32 | 36 | 40 | 44 | 48 | 52 | | |
| Written Informed Consent 4 | Х | | | | | | | | | | | | | | | | |
| Demography | | Х | | | | | | | | | | | | | | | |
| Medical History | | Х | | | | | | | | | | | | | | | |
| SLE History | | Х | | | | | | | | | | | | | | | |
| Therapy History | | Х | | | | | | | | | | | | | | | |
| Physical Examination | | Х | | | | | | | | | | | | | | | |
| Inclusion/Exclusion | | Х | | | | | | | | | | | | | | | |
| Efficacy Assessments | | | | | | | | | | | | | | | | | |
| DAS: SS, SLE Flare Index, PGA <sup>5</sup> | X 1 | Χ | Χ | Χ | Χ | Χ | Х | Χ | Χ | Χ | Χ | Х | Χ | Χ | Х | | |
| SLICC/ACR Damage Index | | Х | | | | | | Х | | | | | | | Х | | |
| Safety Assessments | | | • | • | • | | | | | | | • | | • | • | | |
| Vital Signs <sup>6</sup> | | Χ | Х | Х | Х | Χ | Χ | Χ | Χ | Χ | Х | Χ | Χ | Χ | Х | Χ | |
| Weight, height 6,7 | | Χ | Х | Х | Х | Х | Χ | Χ | Х | Χ | Х | Χ | Χ | Χ | Х | | |
| Symptom-driven Physical Exam | | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | |
| Record Concurrent<br>Medications | | Χ | Х | Х | Х | Х | Х | Χ | Х | Χ | Х | Х | Χ | Х | Х | Х | |
| Adverse Events | | Х | Х | Х | Х | Х | Χ | Х | Х | Х | Х | Х | Χ | Х | Х | Х | |
| Laboratory Assessments | | • | • | | • | • | | | • | | • | | • | • | | | |
| Haematology & Modified<br>Chem 20 (non-fasting) <sup>6</sup> | X | Χ | Х | Х | Х | Х | Х | Χ | Х | Χ | Х | Х | Χ | Х | Х | Х | |
| Urinalysis | Х | Χ | Х | Х | Х | Х | Χ | Χ | Х | Χ | Х | Χ | Χ | Х | Х | Χ | |
| Spot urine (protein to | Х | Χ | Х | Х | Х | Х | Χ | Χ | Х | Χ | Х | Χ | Χ | Χ | Х | | |

| | Screen | | | | | | Ti | reatmen | t Holida | y Study | , | | | | | Follo | w-up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | | |
| Study Day | Up to | 0 <sup>2</sup> | 28 | 56 | 84 | 112 | 140± | 168 | 196± | 224 | 252 | 280± | 308 | 336 | 364 ±7d or | 16-wk | 6 mo |
| J J | -30 ¹ | | ±7d | ±7d | ±7d | ±7d | 7d | ±7d | 7d | ±7d | ±7d | 7d | ±7d | ±7d | Exit | ±7d <sup>3</sup> | ±7d |
| Study Week | | 0 | 4 | 8 | 12 | 16 | 20 | 24 | 28 | 32 | 36 | 40 | 44 | 48 | 52 | | |
| creatinine ratio) 8 | | | | | | | | | | | | | | | | | |
| Pregnancy Test 6, 9 | U | U | U | U | U | U | U | U | U | U | U | U | U | U | U | U | |
| Pharmacogenetic Sampling 10 | | Χ | | | | | | | | | | | | | | | |
| aCL Autoantibody | | Χ | | | | | | | | | | | | | Х | | |
| C3/C4 | Χ | Χ | Χ | Χ | Х | Χ | Χ | Χ | Χ | Χ | Х | Χ | Χ | Χ | Х | | |
| Anti-dsDNA Autoantibodies | Χ | Х | Х | Х | Х | Х | Х | Χ | Х | Х | Х | Х | Х | Х | Х | | |
| ANA Autoantibodies | | Х | | | | | | Χ | | | | | | | Х | | |
| IgG, IgA & IgM 11 | | Х | | Х | | Х | | Χ | | Х | | Х | | Х | Х | | |
| PT/ PTT | | Х | | | | | | | | | | | | | | | |
| Exploratory Lab Assessments | ; | | | | | | | | | | - | | | | | | |
| Pharmacokinetic Sampling 12 | | Χ | | Х | | Х | | X 12 | | Χ | | | | | X 12 | | |
| Immunogenicity 6, 13 | | Х | | | Х | | X 13 | Χ | | | Х | | | | Х | Χ | X 13 |
| BLyS Protein 14 | | | | | | Χ | | Χ | | Χ | | | | | | | |
| B cell Markers <sup>15</sup> | | Х | | Х | | Х | | Χ | | Х | | Х | | | Х | | Х |
| Investigational Product (IP) | | | | | | | | | | | | | | | | | |
| IP Administration 16 | | Х | Х | Х | Х | Х | Х | Χ | Х | Х | Х | Х | Х | Х | <u>X</u> | | |

- 1. DAS = disease activity scales; SS = SELENA SLEDAI; SLE = systemic Lupus Erythematosus; PGA = Physician's Global Assessment; SLICC/ACR = Systemic Lupus International Collaborating Clinics/American College of Rheumatology; ALT = alanine aminotransaminase; AST = aspartate aminotransaminase; PT/PTT = prothrombin time/partial thromboplastin time; BlyS = B Lymphocyte Stimulator; IP = investigational product; aCL = anticardiolipin
- 2. A screening visit of up to 30 days prior to the Day 0 visit will be scheduled for subjects in the treatment holiday and control groups for assessment of SELENA SLEDAI score to assess eligibility.
- 3. The EXIT Visit in the respective feeder continuation studies will serve as the Day 0 visit for all 3 subject groups in this study. Assessments covered for both this study at Day 0 and the Exit visit of the feeder continuation studies need only be performed once and recorded in the appropriate case report forms for each study. Subjects in the control group must be able to receive the 1st dose of belimumab on Day 0 of this study on average 4 weeks (minimum of 2 weeks, maximum of 8 weeks) after the last dose in the feeder continuation study.
- 4. The 16 week follow-up visit will occur at approximately 16 weeks after last dose of investigational product for subjects in the control group who withdraw at any time during the study, or for subjects in the treatment holiday group who withdraw from the study from Week 24 onwards (Visit 7) during the belimumab re-introduction period. The 16-week and 6 month follow-up visits do not apply to subjects in the long-term discontinuation group.
- 5. Obtain written informed consent to participate in this study at the Screening visit.

- 6. Guidelines for scoring proteinuria for SELENA SLEDAI are provided in protocol Section 6.3.1.1.
- 7. Complete assessment prior to belimumab dosing for subjects in the control group (to Week 48) and for subjects in the treatment holiday group (during Weeks 24 to 48 or earlier in the event of a flare). Immunogenicity testing includes quantifying the amount of belimumab present in the samples using the belimumab PK assay.
- 8. For any subject whose weight changes by more than 5% from that recorded at Day 0, use the weight at the current visit for calculating the belimumab dose to be administered. Height measured only at Day 0.
- 9. A 24-hour urine may be done as an additional assessment if clinically indicated (e.g., renal flare).
- 10. Urine pregnancy test results for women of child-bearing potential must be available prior to dosing (during Weeks 0 to 48 in the control group and during Weeks 24 to 48 or earlier in the event of a flare in the treatment holiday group). Can be performed at any time during the visit for females of child-bearing potential in the long-term discontinuation group.
- 11. PGx sampling from consenting subjects recruited from all studies except from study BEL114333. PGx informed consent must be obtained prior to sampling.
- 12. Serum immunoglobulin isotypes: IgG, IgM, IgA.
- 13. Pharmacokinetic sampling at select sites for subjects in the control and treatment holiday groups; subjects in the treatment holiday group can have PK sampling performed at any time during the visit between Weeks 0 and 16. Otherwise, if on a dosing day, sampling must be performed **prior** to dosing. Collect blood samples pre-dose and post-dose at the end of the infusion at Weeks 24 and 52 (or earlier if belimumab is re-started before Week 24 in the event of a severe flare by using the escape option). Subjects in the long-term discontinuation group will have one PK sampling performed at any time during the visit between Weeks 0 and 24. PK sampling for the long-term discontinuation group is not performed after Week 24. Long-term discontinuation subjects withdrawing before Week 24 will have one PK sampling performed at any time during the EXIT visit. PK sampling for long-term discontinuation subjects withdrawing after Week 24 is not performed at the EXIT visit.
- 14. Blood sample for immunogenicity will be taken at Weeks 12, 24, 36 and 52 for all three groups. In addition, a blood sample for immunogenicity will also be taken 4 weeks prior to the reintroduction of belimumab (at Week 20 since belimumab will be reintroduced at Week 24) in the treatment holiday group. A blood sample for immunogenicity must be taken at least 6 months after the final dose of investigational product for any subjects in the control group or treatment holiday group who had an anti-belimumab antibody response at the 16-week follow-up visit (or at the last immunogenicity assessment if 16-week follow-up is not available). Note that serum samples for immunogenicity must be collected pre-dose at the time of dosing from subjects in the treatment holiday group who experience a severe flare prior to Week 24 and consequently receive open-label belimumab as rescue. Immunogenicity blood sample will not be collected at the 6-month follow up visit for subjects in the long-term discontinuation group as this visit does not apply to this subject group.
- 15. Measured in treatment holiday group at Weeks 16 and pre-dose at Week 24. Measured in long-term discontinuation group at Weeks 16, 24 and 32. Not measured in control group.
- 16. Biological Markers include FACS of peripheral lymphocytes: B lymphocytes (CD20+, CD20+/27+ memory, CD20+/27- naïve, CD20+/69+ activated, CD20+/138+ plasmacytoid, CD19+/27BRIGHT/38BRIGHT SLE subset and CD20-/138+ plasma cells). Note: B cell markers will not be collected at the 6-month follow up visit for subjects in the long-term discontinuation group as this visit does not apply to this subject group.
- 17. Only subjects in the control group will receive belimumab 10 mg/kg during Weeks 0 through 20 inclusive; subjects in the control group must be able to receive the **first** dose of belimumab **in this study** 4 weeks (minimum of 2 weeks, maximum of 8 weeks) after the last dose in their **previous** open-label continuation study. Subjects in the control group and treatment holiday groups will receive belimumab from Weeks 24 through 48 although subjects in the treatment holiday group may be treated with belimumab **prior** to Week 24 as determined by the investigator in the event of increased SLE activity. When belimumab therapy is re-started, subjects in the treatment holiday group will remain under clinical supervision for 3 hours after completion of the first 2 infusions. At the **Week 52** visit, only subjects in the treatment holiday and control groups who are continuing belimumab therapy beyond this time will be dosed.

# 13.2.3. Time and Events Table (Additional Years)

| Study Visit (Weeks) 1 | 4 | 8 | 12 | 16 | 20 | 24 | 28 | 32 | 36 | 40 | 44 | 48 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Day | 28<br>±7d | 56<br>±7d | 84<br>±7d | 112<br>±7d | 140<br>±7d | 168<br>±7d | 196<br>±7d | 224<br>±7d | 252<br>±7d | 280<br>±7d | 308<br>±7d | 336<br>±7d |
| Efficacy Assessments | | | | | | | | | | | | |
| Disease Activity Scales: SELENA SLEDAI,<br>SLE Flare Index, and PGA <sup>2</sup> | | | | | | Х | | | | | | Х |
| SLICC/ACR Damage Index | | | | | | | | | | | | Χ |
| Safety Assessments | | | | | | | | | | | | |
| Symptom-driven Physical Exam | | | | | | Х | | | | | | Χ |
| Record Concurrent Medications | Χ | Х | Χ | Х | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ |
| Adverse Events | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ |
| Vital Signs <sup>3, 4</sup> | Χ | Χ | Χ | Χ | Х | Х | X | X | Χ | Χ | Χ | Χ |
| Laboratory Assessments | | | | | | | | | | | | |
| Haematology & Modified Chem 20 (non-fasting) 3, 5 | | | | | | Х | | | | | | Х |
| Urinalysis 5, 6 | | | | | | Χ | | | | | | Χ |
| Spot urine (protein to creatinine ratio) 3, 5, 6 | | | | | | Х | | | | | | Χ |
| Urine Pregnancy Test 3, 5, 7 | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ |
| C3, C4, Anti-dsDNA Autoantibodies 3, 5 | | | | | | Χ | | | | | | Χ |
| IgG <sup>3, 5, 8</sup> | | | | | | | | | | | | Χ |
| IgA & IgM <sup>3, 5, 8</sup> | | | | | | | | | | | | Χ |
| Exploratory Lab Assessments | | | | | | | | | | | | |
| Immunogenicity <sup>3,9</sup> | | | | | | Х | | | | | | Χ |
| B cell Markers <sup>10</sup> | | | | | | | | | | | | Χ |
| Investigational Product | | | | | | | | | | | | |
| Belimumab Administration 4, 11 | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ |

- 1. Calendar represents a yearly (48-week) ongoing visit schedule until the subject is terminated from the study.
- Guidelines for scoring proteinuria for SELENA SLEDAI are provided in protocol Section 6.3.1.1.
- 3. Assessments performed prior to dosing.
- 4. For any subject whose weight changes by more than 5% from that recorded at Day 0, use the weight at the current visit for calculating the belimumab dose to be administered.
- 5. During "Additional years", investigators can obtain any of the same laboratory assessments that are mentioned for Year 1 (haematology, modified Chem 20, urinalysis, spot urine to creatinine ratio, urine pregnancy, C3, C4, anti-ds DNA autoantibodies, IgG, IgA, and IgM), as unscheduled laboratory tests at any time during Year 2 and beyond, if clinically indicated. Any additional laboratory tests beyond this, if not related to the protocol, will be the responsibility of the investigator and subject.
- 6. A 24-hour urine may be done as an additional assessment if clinically indicated (e.g., renal flare).
- 7. Results of urine pregnancy tests in women of child-bearing potential must be available prior to belimumab dosing.
- 8. Serum immunoglobulin isotypes: IgG, IgM, IgA.
- 9. Immunogenicity testing includes quantifying the amount of belimumab present in the samples using the belimumab PK assay.
- 10. Biological Markers include FACS of peripheral lymphocytes: B lymphocytes (CD20+, CD20+/27+ memory, CD20+/27- naïve, CD20+/69+ activated, CD20+/138+ plasmacytoid, CD19+/27BRIGHT/38BRIGHT SLE subset and CD20-/138+ plasma cells).
- 11. After completion of the Week 48 visit during year 1 of the study, subjects in the treatment holiday and control groups can continue to receive belimumab therapy at 4-weekly intervals in the maintenance phase of this study. Subjects who withdraw from belimumab therapy during this maintenance phase will complete the Exit and follow-up visits detailed in the Year 1 Time and Events Table. The Exit visit Schedule should be scheduled 4 weeks after the final belimumab dose and the 16-week follow-up visit 16 weeks after the final belimumab dose.

## 13.3. Appendix 3: Assessment Windows

# 13.3.1. Mapping of the Maintenance Phase Visits for Subjects with an Escape Visit

In the eCRF, the next visit provided following the Escape visit is the Year 2 Week 8 visit, when chronologically the next visit would be the Year 2 Week 4 visit. Therefore, the maintenance phase visits for subjects with an Escape visit will be re-mapped in the ADaM analysis data sets to the maintenance phase visit, so that the visits align chronologically with those for subjects who complete the 52-week treatment phase and subsequently enter the maintenance phase.

If an Escape visit is present, mapping will occur as follows:

| | SDTM Variable | ADAM Variable |
|---|---|---|
| Domain | VISITNUM<br>VISIT | AVISITN<br>AVISIT |
| All | 190<br>ESCAPE | 190<br>ESCAPE |
| All | 220<br>YEAR 2 WEEK 8 | 210<br>YEAR 2 WEEK 4 |
| All | 230<br>YEAR 2 WEEK 12 | 220<br>YEAR 2 WEEK 8 |
| All | 240<br>YEAR 2 WEEK 16 | 230<br>YEAR 2 WEEK 12 |
| The mapping will continue in this pattern for subsequent visits. | | |

## 13.3.2. Mapping of Week 16 and 6-month Follow-up Visits

The 16-week and 6-month follow-up visits will be re-mapped in the ADaM analysis data sets so that they sort in chronological sequence when using the numeric visit number.

| | SDTM Variable | ADAM Variable |
|--------|------------------------|-------------------------|
| Domain | VISITNUM<br>VISIT | AVISITN<br>AVISIT |
| All | 170<br>16 WK FOLLOW-UP | 9100<br>16 WK FOLLOW-UP |
| All | 180<br>6 MO FOLLOW-UP | 9200<br>6 MO FOLLOW-UP |

## 13.3.3. Analysis Visit and Analysis Visit Number

The data are analyzed according to the planned visit assignment in the data.

Exit/withdrawal visits must be slotted to the appropriate planned visit according to the study phase. This will only be done for subjects that withdrew early and did not complete the 52-week treatment phase. Unscheduled laboratory visits will also be slotted to the appropriate planned visit.

The Analysis Visit is assigned based on the interval in which the Study Day for the exit/withdrawal visit or unscheduled laboratory visit falls according to intervals (inclusive) provided below. For completeness, the table also includes visits which are not slotted; these visits will have 'na' for 'not available' listed for the Interval Start and End Day.

| | Analysis | | Interval Start Day | Interval End Day |
|---|---|---|---|---|
| <b>Analysis Visit</b> | Visit Number | Target Study Day <sup>1</sup> | - | _ |
| Screening | 10 | -34 | na | na |
| 52-week Treatment | Phase visits: | | | |
| Baseline | 20 | 1 | na | na |
| Week 4 | 30 | 29 | 22 | 42 |
| Week 8 | 40 | 57 | 43 | 70 |
| Week 12 | 50 | 85 | 71 | 98 |
| Week 16 | 60 | 113 | 99 | 126 |
| Week 20 | 70 | 141 | 127 | 154 |
| Week 24 | 80 | 169 | 155 | 182 |
| Week 28 | 90 | 197 | 183 | 210 |
| Week 32 | 100 | 225 | 211 | 238 |
| Week 36 | 110 | 253 | 239 | 266 |
| Week 40 | 120 | 281 | 267 | 294 |
| Week 44 | 130 | 309 | 295 | 322 |
| Week 48 | 140 | 337 | 323 | 350 |
| Week 52 | 150 | 365 | 351 | 378 |

| | Analysis | | Interval Start Day | Interval End Day |
|---|---|---|---|---|
| Analysis Visit | Visit Number | Target Study Day <sup>1</sup> | | |
| <sup>1</sup> Day 0 visit date in s | tudy 116027 = S | tudy Day 1. | | |

# 13.3.4. Windows for Assessment of Post-injection/infusion sensitivity reactions (PISR) and hypersensitivity reactions (HSR)

The windows for assessment of PISR/HSR, as described in the AESI definitions in Section 13.9.2, are as follows:

| Date of Infusion | | |
|---|---|---|
| Day 1 | Day 2 | Day 3 |
| SMQ narrow, broad and algorithmic searches (On day of injection/infusion or within 3 | | |
| days of injection/infusion) | | |

# 13.4. Appendix 4: Study Phases and Treatment Emergent Adverse Events

#### 13.4.1. Treatment Phases

- Visits, assessments and events will be classified according to the time of occurrence relative to the following cut-point dates for each treatment group.
- For convenience and ease of data presentation, the 52-Week Treatment Phase has the same name designation for all three treatment groups, even though the LTC group does not receive treatment at all during this phase and the TH group receives treatment for only the second half of the phase.
- Only the TC and TH groups are eligible to participate in the Maintenance Phase.
- If an AE start date falls on the Day 0 date, then it will be considered treatment emergent (i.e., fall in the 52-week treatment phase). If a concomitant medication start date falls on the Day 0 visit date, the concomitant medication will be considered to fall in the 52-week treatment phase. Any other assessments that fall on the Day 0 visit date will be considered to occur in the pre-study phase.
- For the TC group, if the first infusion date differs from the Day 0 visit date, then the first infusion date will be used as the phase cut-point.
- Other than Day 0, if an assessment or event occurs on the same date as a phase cutpoint, then the event will be considered to fall in the previous phase. For example, if a new prednisone dose starts on the same date as the Week 24 visit date and then continues for a total of 7 days, then the first day of that prednisone dose will fall into the Holiday Phase and the remaining 6 will fall into the Re-start phase.
- For AEs, if the AE Onset date is missing, then the AE will be considered to occur in the 52-week treatment phase.
- For the TH group, a subject who re-starts treatment prior to Week 24 will not have a Re-Start phase.

## 13.4.1.1. Treatment Holiday Group

| Endpoint | Day 0 Visit<br>Parent<br>Study | Day 0 Visit<br>BEL116027<br>Study | Week 24/<br>TX Re-start<br>Visit | Week 52/<br>Exit/Escape<br>Visit | Week<br>16<br>Follow-<br>up Visit |
|---|---|---|---|---|---|
| | Baseline | | | | |
| Flare, PGA, Prednisone, | <b>N</b> 1/A | 52-Week Trea | atment Phase | Maintenance | N1/A |
| SLICC | N/A | Holiday Phase | Re-start Phase | Phase | N/A |
| Baseline | | | | | |
| SS, Auto-antibodies | Pre-Study | 52-Week Trea | atment Phase | Maintenance | N/A |
| Immunoglobulins,<br>B-cells [1], BLyS | Phase | Holiday Phase | Re-start Phase | Phase | IN/A |
| | | Baseline | | | • |
| Rebound [2] | Pre-Study | 52-Week Trea | atment Phase | NI/A | N/A |
| | Phase | Holiday Phase | N/A | N/A | IN/A |
| | | Baseline | | | |
| Adverse Events, Lab | NI/A | 52-Week Trea | atment Phase | Maintenance | 21/2 |
| Parameters, Vital Signs, Con<br>Meds Immunogenicity [1] | N/A | Holiday Phase | Re-start Phase | Phase | N/A |

N/A = Not Applicable.

<sup>[1]</sup> Immunogenicity and B-cells may also be collected at the 6-month follow-up visit. The 6-month follow-up visit is not represented in the diagram since it does not define a treatment phase of the study.

<sup>[2]</sup> Rebound is only assessed up to the Week 24/Treatment re-start visit.

## 13.4.1.2. Treatment Control Group

| Endpoint | Day 0 Visit<br>Parent Study | Day 0 Visit<br>BEL116027<br>Study [1] | Week 24 Visit | Week 52/<br>Exit Visit | Week<br>16<br>Follow<br>-up<br>Visit |
|---|---|---|---|---|---|
| Baseline | | | | | |
| Flare, PGA, Prednisone, SLICC | N/A | 52-Week Trea | Maintenance<br>Phase | N/A | |
| Baseline | | | | | |
| SS, Auto-antibodies<br>Immunoglobulins,<br>B-cells [2], BLyS | Pre-Study<br>Phase | 52-Week Trea | atment Phase | Maintenance<br>Phase | N/A |
| | | Baseline | | | |
| Rebound [3] | | 52-Week Trea | atment Phase | | |
| | Pre-Study<br>Phase | First 24 Weeks | N/A | N/A | N/A |
| | | Baseline | | | |
| Adverse Events, Lab<br>Parameters, Vital Signs, Con<br>Meds , Immunogenicity [2] | N/A | 52-Week Trea | atment Phase | Maintenance<br>Phase | N/A |

N/A = Not Applicable.

<sup>[1]</sup> If the first infusion date differs from the Day 0 visit date, then the first infusion date will be used as the phase cut-point.

<sup>[2]</sup> Immunogenicity and B-cells may also be collected at the 6-month follow-up visit. The 6-month follow-up visit is not represented in the diagram since it does not define a treatment phase of the study.

<sup>[3]</sup> Rebound is only assessed up to the Week 24 visit.

## 13.4.1.3. Long-term Discontinuation Group

| Endpoint | Day 0 Visit<br>Parent<br>Study | Day 0 Visit<br>BEL116027 Study | BEL116027 Study | | Week 52/<br>Exit Visit | |
|---|---|---|---|---|---|---|
| | - | Baseline | | | | |
| Flare, PGA, Prednisone, SLICC | N/A | N/A | 52-Week 7<br>Pha | | N/A | |
| | | Baseline | • | | | |
| SS, Auto-antibodies<br>Immunoglobulins, BLyS | N/A | Pre-Study Phase | 52-Week Treatment<br>Phase | | | N/A |
| | | Baseline | • | | | |
| Rebound | N/A | Dro Ctudy Phono | 52-Week 7<br>Pha | N1/A | | |
| | IN/A | Pre-Study Phase | First 24<br>Weeks | N/A | N/A | |
| | | Baseline | | | | |
| Adverse Events, Lab<br>Parameters, Vital Signs,<br>Con Meds | N/A | N/A | 52-Week Treatment<br>Phase | | N/A | |

N/A = Not Applicable.

| Treatment<br>State | Treatment<br>Group | Definition |
|---|---|---|
| Treatment<br>Emergent | TH, LTD | AE Onset Date ≥ Day 0 visit date |
| Treatment<br>Emergent | TC | AE Onset Date ≥ Date of First Infusion in BEL116027 |
| Onset Time<br>Since 1st<br>Dose (Days) | TH, TC | If Date of First Infusion in BEL116027> AE Onset Date: = AE Onset Date - Date of First Infusion in BEL116027 If Date of First Infusion in BEL116027≤ AE Onset Date = AE Onset Date - Date of First Infusion in BEL116027+1 =Missing otherwise. |
| Onset Time<br>Since Study<br>Start (Days) | TH, TC, LTD | If Day 0 visit date > AE Onset Date: = AE Onset Date – Day 0 visit date If Day 0 visit date ≤ AE Onset Date = AE Onset Date - Day 0 visit date +1 =Missing otherwise. |
| Duration<br>(Days) | TH, TC, LTD | AE Resolution Date – AE Onset Date + 1 |
| Drug-related | TH, TC, LTD | If relationship is marked 'YES' on Inform/CRF OR value is missing. |

## 1. NOTES:

• If the AE Onset date is missing, then the AE will be considered as treatment emergent.

# 13.5. Appendix 5: Data Display Standards & Handling Conventions

## 13.5.1. Reporting Process

| Software | |
|---|---|
| The currently supported versions of SAS software will be used. | |
| Reporting Area | |
| HARP Server | US1SALX00259 |
| HARP Compound and Reporting effort | GSK1550188/BEL116027/final_01 |
| Analysis Datasets | |
| <ul> <li>Analysis datasets will be created according to CDISC standards (SDTM IG Version 3.2 &amp; ADaM IG<br/>Version 1.0).</li> </ul> | |
| Generation of RTF Files | |
| RTF files will be generated for all tables in the final_cdisc RE | |

## 13.5.2. Reporting Standards

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated (IDSL Standards Location: https://spope.gsk.com/sites/IDSLLibrary/SitePages/Home.aspx):
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics
- Do not include subject level listings in the main body of the GSK Clinical Study Report. All subject level listings should be located in the modular appendices as ICH or non-ICH listings

#### **Formats**

- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected, unless otherwise stated.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses:
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days
    on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study agent dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.

#### **Unscheduled Visits**

- Unscheduled visits will not be included in summary tables.
- Unscheduled visits will be included in figures unless their inclusion contributes adversely to

| visual presentation or interpretation of the figure. | |
|---|---|
| All unscheduled v | All unscheduled visits will be included in listings. |
| Descriptive Summary Statistics | |
| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data | N, n, frequency, % |
| Graphical Displays | |
| Refer to IDSL Statistical Principals 7.01 to 7.13. | |

# 13.5.3. Reporting Standards for Pharmacokinetic

| Pharmacokinetic Concentration Data | |
|---|---|
| Descriptive<br>Summary Statistics<br>(Log Transformed) | N, n, geometric mean, 95% CI of geometric mean, standard deviation (SD) of log transformed data and between geometric coefficient of variation (CVb (%)) will be reported. $ \text{CV}_{\text{b}} \text{ (\%)} = \sqrt{\left(\text{exp}(\text{SD}^2) - 1\right) * 100} $ (SD = SD of log transformed data) |
| Parameters Not<br>Being Log<br>Transformed | N, n mean, 95% CI, standard deviation (SD), median, 25 <sup>th</sup> and 75 <sup>th</sup> percentile, minimum and maximum will be reported. |
| Pharmacokinetic Parameter Data | |
| Is NQ impacted PK<br>Parameters Rule<br>Being Followed | Yes, refer to Standards for Handling NQ Impacted PK Parameters |

## 13.6. Appendix 6: Derived and Transformed Data

#### 13.6.1. General

## **Multiple Measurements at One Time Point**

- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- Subjects having both High and Low values for Normal Ranges at any post-baseline visits for safety parameters will be counted in both the High and Low categories of "Any visit postbaseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.

## **Study Day**

- Calculated as the number of days from the Day 0 Visit Date (i.e., Day 1) to the assessment date or visit date of interest (Ref Date)
  - Ref Date = Missing → Study Day = Missing
  - Ref Date < Day 0 Visit Date → Study Day = Ref Date Day 0 Visit Date</li>
  - Ref Data ≥Day 0 Visit Date → Study Day = Ref Date –Day 0 Visit Date + 1

## 13.6.2. Study Population

## **Demographics**

## **Study Phases Definitions for Disposition**

- Completion/withdrawal for the 52-Week Treatment Phase will be derived as follows:
  - Withdrawn if the subject completion status is marked as No and the subject has no visits during the maintenance phase.
  - Complete if the subject completion status is marked as Yes and the subject has no visits during the maintenance phase.
- Completion/withdrawal for the Maintenance Phase will be derived as follows:
  - Withdrawn if the subject completion status is marked as No and the subject has at least one visit during the maintenance phase.
  - Complete if the subject completion status is marked as Yes and the subject has at least one visit during the maintenance phase.

#### Age

- GSK standard IDSL algorithms will be used for calculating age where birth date will be imputed as follows:
  - Any subject with a missing day will have this imputed as day '15'.
  - Any subject with a missing date and month will have this imputed as '30th June'.
- Birth date will be presented in listings as 'YYYY'.
- Analysis age is derived in years relative to the Day 0 visit date, and is calculated in SAS as follows:

Analysis Age (years) INTCK('year', Date of Birth, Day 0 Date)

- ( MONTH(Day 0 Date) < MONTH(Date of Birth)

| Dam | | - n h | |
|-----|------|-------|-----|
| Dem | ogra | apn | ICS |

or (MONTH(Day 0 Date) eq MONTH(Date of Birth)

and DAY(Day 0 Date) < DAY(Date of Birth) )

#### **Proteinuria**

- For analysis, urine protein in g/24-hour will be approximated by the urine protein:creatinine ratio (uPCR).
- The value for reporting and analysis is stored in the uPCR result variable corresponding to the
  original unit in the SI dataset. Depending on the study, units for uPCR may be reported in g/g or
  mg/mg. As long as the units are the same in the numerator and denominator, the ratio will be
  the same.
- The SI dataset standard unit is reported in mg/mmol is not used for reporting and analysis purposes in this study.

## **Concomitant medications**

- Concomitant medications are defined as
  - a. Medications that start on or before the Day 0 visit date and end on or after the Day 0 visit date. or
  - b. Medications that start after the Day 0 visit date
- Medications that meet criterion 'a' are considered to be in use at baseline.
- Medications will be assigned to the 52-week treatment or maintenance phases, as per the definitions in Section 13.4.1.
- Medications with partial or missing start and/or stop dates will be assumed to be concomitant
  unless there is evidence through comparison of partial dates to suggest otherwise, for example
  if the day is missing, then the month and year will be compared to the month and year of the
  first dose date of study treatment and if the month and year are the same or later, then the
  medication will be considered concomitant.

#### Allowable SLE Medications at Baseline

There are 5 medication categories that are evaluated. These medication categories are defined in the table below and stored in the variable CMSCAT. Only medications providing systemic exposure are evaluated. Systemic exposure is based on the route of administration. A flag variable for systemic exposure when CMSCAT is not blank is defined below and stored in the variable SYSTEMIC. The medication must have one of the defined medication categories below (CMSCAT ne blank) and must provide systemic exposure (SYSTEMIC='Y').

| Medication Category (CMSCAT) | Rule |
|---|---|
| Anti-malarials | Set CMSCAT to "ANTIMALARIALS" if the preferred |
| | term begins with "QUINACRINE", "QUININE", |
| | "HYDROXYCHLOROQUINE", |
| | "MEPACRINE", or "CHLOROQUINE" |
| Steroids | Set CMSCAT to 'STEROIDS' if at least one |
| | associated ATC code (ATCCD1 – ATCCD6) begins |
| | with 'H02' |

| CMSCAT to 'IMMUNOSUPPRESSANTS' if at tone associated ATC code (ATCCD1 – CD6) begins with 'L04A' or the preferred term ns with "CYCLOPHOSPHAMIDE" or RCAPTOPURINE". CMSCAT to NSAIDs if at least one associated code (ATCCD1 – ATCCD6) begins with 'M01A'. CMSCAT to "ASPIRIN" if CMDECOD contains ETYLSALICYLIC ACID" or |
|---|
| code (ATCCD1 – ATCCD6) begins with 'M01A'. CMSCAT to "ASPIRIN" if CMDECOD contains |
| CMSCAT to "ASPIRIN" if CMDECOD contains |
| ETYLSALICYLATE LYSINE". |
| to "PROHIBITED" if any of following conditions are met, if CMDECOD als "INVESTIGATIONAL DRUG", MUNOGLOBULIN", ALIMUMAB", "ETANERCEPT", "INFLIXIMAB", "UXIMAB", "ABATACEPT", "ANAKINRA", LIMUMAB", "CERTOLIZUMAB" for view of the surgeries/procedures form indicates subject had "PLASMAPHERESIS". |
| se medications will be identified based on a cal review of all the concomitant medications gned the following drug collection codes in the 37301, 50192401, 53020201, 53060901, 56001, 53927401, 53959101, 53959201, 50601, 54619401, 54731901, 54908201, 54101 |
| ) |
| MSCAT=blank |
| CMSCAT ne blank and the route of |

## **Treatment Compliance**

• Treatment compliance for patients completing the 52 week treatment phase or withdrawals is calculated as:

treatment compliance (%)

= 100 
$$imes rac{Number\ of\ infusions\ prescribed-Number\ of\ infusions\ missed}{Number\ of\ infusions\ prescribed}$$

- Prescribed number of infusions will be 7 for the TH arm and 13 for the TC arm, except for TH subjects who escape to the Maintenance Phase. For TH subjects who escape, the treatment compliance will be missing. The Week 52 infusion is considered to be the first infusion of the maintenance phase.
- NB: for withdrawals the number of infusions prescribed is the number from Day 0 up to the withdrawal date

## **Extent of Exposure**

- Number of days of exposure to study treatment during the 52-week Treatment Phase will be calculated based on the formula:
  - Duration of Exposure in Days = (Date of last infusion in BEL116027 52-week treatment Phase—Date of first infusion in BEL116027) + 28
- The Week 52 infusion is considered to be the first infusion in the Maintenance Phase, and will
  not be considered in this calculation.
- Subjects who were enrolled in the TH and TC groups but did not receive an infusion will be categorised as having zero days of exposure.
- Exposure will not be calculated for the LTD group.
- Only complete dates will be used when calculating duration of exposure.
- Exposure will not be adjusted for skipped infusions.

## 13.6.3. **Efficacy**

## SLE Flares and Severe Flares, and Renal Flares

#### **Baseline Flares**

• Baseline flares will be summarized using the data from the eCRF SFI data collection for the Day 0 visit. Per eCRF completion guidelines, the data collected at the Day 0 visit represents the flare data since the previous visit (i.e. the last visit in the feeder continuation study).

## **SLE Flares and Severe SLE Flares**

| SLE Flares and Severe Flares, and Renal Flares |
|---|
| CCI - This section contained Clinical Outcome Assessment data collection questionnaires or indices, which are protected by third party copyright laws and therefore have been excluded. |
| unitu party copyright laws and therefore have been excluded. |

- SFI reports the first mild /moderate or severe flare occurrence since the last visit assessment.
- The SLEDAI criteria will be assessed programmatically to determine if the SELENA SLEDAI criteria for a flare has been met and used for the assessment of flare, irrespective of what was recorded on the SFI form.
- Although there are boxes on the form for the investigator to classify the most recent flare to mild/moderate or severe, the classification will be re-derived from the subcategory scores. Flares originally marked severe will be downgraded to "Not Severe" if the only reason marked is a change in SELENA SLEDAI score to > 12.
- In this case, if any of the mild/moderate reasons are checked or if the modified SELENA SLEDAI score has a change from previous visit of at least 3, then the flare will be considered Mild/Moderate.
- Flares that are marked mild/moderate where the only reason checked is SELENA SLEDAI increase of at least 3 points but not more than 12 points will be re-derived using the modified SELENA SLEDAI score.
- If it's found that the change is not actually  $\geq 3$ , and no other reasons are checked,

## SLE Flares and Severe Flares, and Renal Flares

then the flare will not be counted.

## **Renal Flares**

A SLE Renal flare is defined as the occurrence of at least 1 or more of the following in 2 or more consecutive visits during the study. (NB: at least 1 of the same criteria must be present on at least 2 consecutive visits)

Increased Proteinuria (using spot urine)

A reproducible increase in 24-hour urine protein levels (as measured in uPCR) to:

• >1g if the baseline (Day 0)value was <0.2g

OR

• >2g if the baseline (Day 0) value was between 0.2g and 1g

OR

• More than twice the value at baseline (Day 0) if the baseline value (Day 0)was >1g

## Impaired Renal Function

- A reproducible decrease in GFR of >20%, accompanied by proteinuria (>1), and/or cellular (RBC and WBC) casts.
- [Alarcón-Segovia, 2003].

GFR is estimated by the Cockcroft-Gault equation [Cockcroft, 1976] for creatinine clearance in mL/min.

## Cockeroft-Gault Equation

| Cl <sub>cr</sub> (mL/min) = | (140-age (yrs)) x weight (kg)<br>x 0.85 if fema | |
|---|---|---|
| | 72 x serum creatinine (mg/dL) | _ |

<sup>&</sup>quot;Reproducible" requires the criterion to be met at two consecutive visits, including unscheduled visits.

The following table identifies the lab parameters to be used to evaluate the criteria in the renal flare definition above.

| Criterion | Parameter | SI Dataset<br>LBTESTCD |
|---|---|---|
| Proteinuria | Urine Protein:Creatinine Ratio (mg/mg) | PRTCRT_URQ |
| GFR | Creatinine Clearance estimated by the Cockcroft-Gault equation (mL/min) | CRTCE_PLR |
| Cellular casts: | | |
| WBC cellular casts | WBC cellular casts | WBCSTM_URQ |
| dysmorphic RBCs | dysmorphic RBCs | DRBCM_URQ |

## SLE Flares and Severe Flares, and Renal Flares

#### **Derivation for rates of SFI flares**

• Within a treatment group, the unadjusted flare (severe flare) rate per subject-year in a given phase will be calculated as:

Unadjusted flare (severe flare) rate per subject-year =

total number of flares (severe flares) in the phase / total number of years of follow-up time in the phase.

• The calculation will not include baseline flares in the 116027 study.

#### Follow-up time derivation for rates of SFI flares

| Phase | Treatment<br>Group | Definition |
|---|---|---|
| 52-week<br>Treatment<br>Phase | TC, LTD | (Week 52/Exit visit date – Day 0 date + 1)/ 365.25. |
| TH Phase | TH | (Week 24/TX re-start date – Day 0 date + 1)/ 365.25. |
| RS Phase | TH | (Week 52/Exit visit – Week 24/TX re-start date)/ 365.25. |

## **SELENA SLEDAI Organ System Domains**

SELENA SLEDAI assessments consist of 24 individual weighted items in which signs and symptoms, laboratory tests, and physician's assessment for each of 8 organ systems are given a weighted score and summed if present (marked 'Yes') at the time of the visit or in the preceding 10 days. The maximum theoretical score is 105 (all 24 descriptors present simultaneously) with 0 indicating inactive disease (marked 'No'), but in practice few subjects have scores > 45 [Buyon, 2005; Petri, 2005].

Organ system domain scores are the sum of the weights of items within the organ domain as defined in the table below.

In this study, proteinuria is evaluated using spot-urine protein [represented as protein-creatinine ratio or PC Ratio (Add ref to 9.3.13) in the laboratory dataset] in lieu of the 24-hour urine collection. PC ratio in mg/mg is considered equivalent to g/24-hr urine protein.

If the P/C ratio value is missing, then the value from the previous visit will be used. Specifically, the assessment for proteinuria indicated on the CRF will be used to calculate the SELENA SLEDAI score. In the eCRF, laboratory items on the SLEDAI may also be ticked 'unknown' to indicate the lab test was not available. The laboratory items are: urinary casts, hematuria, proteinuria, pyuria, low complement, increased DNA binding, thrombocytopenia, and leukopenia. Responses of 'Unknown' will be managed via LOCF

List of organ systems, items, and weights for the assessments are provided.

| Organ System | Descriptor | Weight |
|----------------------------------|------------------------|--------|
| [1] CNS | Seizure | 8 |
| | Psychosis | 8 |
| | Organic Brain Syndrome | 8 |
| | Visual Disturbance | 8 |
| | Cranial Nerve Disorder | 8 |
| | Lupus Headache | 8 |
| | CVA | 8 |
| [2] Vascular | Vasculitis | 8 |
| [3] Musculoskeletal | Arthritis | 4 |
| | Myositis | 4 |
| [4] Renal | Urinary Casts | 4 |
| | Hematuria | 4 |
| | Proteinuria | 4 |
| | Pyuria | 4 |
| [5] Mucocutaneous | Rash | 2 |
| | Alopecia | 2 |
| | Mucosal Ulcers | 2 |
| [6] Cardiovascular & Respiratory | Pleurisy | 2 |
| | Pericarditis | 2 |
| [7] Immunologic | Low Complement | 2 |
| | Increased DNA Binding | 2 |
| [8] Constitutional | Fever | 1 |
| [9] Hematologic | Thrombocytopenia | 1 |
| | Leukopenia | 1 |

#### **PGA**

- The PGA is collected on a 10cm visual analogue scale (VAS).
- The standard scoring range for the PGA is 0 to 3, and the score will be rescaled for standard reporting by multiplying the collected score by 3/10.
- During study conduct, it was noted that some sites erroneously received PGA scales that were 9.5cm in length due to a printing error, and some subjects utilized these scales before the error was discovered. Per Notes to File (08Jan2015, and 20Sep2017), an evaluation was performed and the decision was taken that this would result in minimal differences and not expected to affect any outcomes, and therefore it was unnecessary to adjust the analysis.

## **Prednisone Equivalent Conversion**

## **Identification of Steroids**

- A concomitant medication is identified as a steroid if
  - At least one associated ATC code (ATCCD1 ATCCD6) begins with 'H02.' AND
  - The route meets the following criteria:
    - Provides systemic exposure: oral, subcutaneous, intramuscular, intradermal, and intravenous.
    - Although not systemic, intra-articular steroids are also identified for

prohibited medication rules.

- Topical routes of administration are excluded (e.g., topical, conjunctival, intranasal).
- Steroid doses will be converted to the prednisone-equivalent dose.
- At data base release, all preferred terms identified with an ATC code beginning with 'H02' will be reviewed to ensure a conversion factor exists for all terms with a systemic or intra-articular route of administration.
- Similarly, all routes of administration for preferred terms with an ATC code beginning with 'H02' will be reviewed to ensure all systemic or intra-articular routes have been identified in the list above.
- In order to be converted, the frequency and dose of the steroid must be present with the unit dose in milligrams (mg).
- Reported dose for systemic steroid is converted to prednisone equivalent dose using conversion factor for each particular medication (refer to online calculator http://www.globalrph.com/corticocalc.htm).
  - Prednisone Equivalent Daily Dose (mg) = Collected Dose (mg) x Conversion Factor x Frequency Factor

## **Average Daily Dose Derivation**

- Average daily prednisone dose at baseline is based on all days from the Screening visit date up to and including the Day 0 visit date.
- Post-baseline, average daily prednisone dose is based on all days between visits including the current visit date.
- Average Daily Dose (mg/day) = Sum of Prednisone Equivalent Daily Dose (mg) across all days in the visit interval / Number of days in the visit interval

| Prednisone Conversion Factors (mg) | |
|------------------------------------|---------------------------------------|
| | Conversion factor for converting to a |
| Preferred term | prednisone-equivalent dose |
| BETAMETHASONE | 8.3333 |
| BETAMETHASONE DIPROPIONATE | 8.3333 |
| BETAMETHASONE SODIUM PHOSPHATE | 8.3333 |
| BETROSPAM | 8.3333 |
| BUDESONIDE | 0.3333 |
| CELESTONA BIFAS | 7.5 |
| CORTISONE | 0.2 |
| CORTISONE ACETATE | 0.2 |
| CRONOLEVEL | 8.3333 |
| DEFLAZACORT | 0.8333 |
| DEPO-MEDROL MED LIDOKAIN | 1.25 |
| DEXAMETHASONE | 6.6667 |
| DEXAMETHASONE ACETATE | 6.6667 |
| DEXAMETHASONE SODIUM PHOSPHATE | 6.6667 |
| FLUOCORTOLONE | 3 |
| HYDROCORTISONE | 0.25 |
| HYDROCORTISONE ACETATE | 0.25 |
| HYDROCORTISONE SODIUM SUCCINATE | 0.25 |
| MEPREDNISONE | 1.25 |
| METHYLPREDNISOLONE | 1.25 |
| METHYLPREDNISOLONE ACETATE | 1.25 |
| METHYLPREDNISOLONE SODIUM | 1.25 |
| SUCCINATE | 20 |
| PARAMETHASONE | 2.5 |
| PREDNISOLONE | 1 |
| PREDNISOLONE ACETATE | 1 |
| PREDNISOLONE SODIUM PHOSPHATE | 1 |
| PREDNISOLONE SODIUM SUCCINATE | 1 |
| PREDNISONE | 1 |
| PREDNISONE ACETATE | 1 |
| TRIAMCINOLONE | 1.25 |
| TRIAMCINOLONE ACETATE | 1.25 |
| TRIAMCINOLONE ACETONIDE | 1.25 |
| Frequency Factors | 1.20 |
| Frequency | Factor |
| BID | 2 |
| BIW | 2/7 |
| OAM | 1/30 |
| Once | 1/30 |
| PRN | null |
| Q2H | 12 |
| Q2W | 1/14 |
| Q3H | 8 |

| Q3MO | 1/84 |
|------------------|------|
| Q3w | 1/21 |
| Q4H | 6 |
| Q4W | 1/28 |
| Q6H | 4 |
| Q8H | 3 |
| QAM | 1 |
| QD | 1 |
| QH | 24 |
| QHS | 1 |
| QID | 4 |
| QOD | 1/2 |
| QPM | 1 |
| QW | 1/7 |
| QWK | 1/7 |
| TID | 3 |
| TIW | 3/7 |
| UNK | null |
| 2 TIMES PER WEEK | 2/7 |
| 3 TIMES PER WEEK | 3/7 |
| EVERY 2 WEEKS | 1/14 |
| EVERY 3 WEEKS | 1/21 |
| EVERY 4 Weeks | 1/28 |
| EVERY WEEK | 1/7 |

## 13.6.4. Safety

#### **Adverse Events**

## **Adverse Events of Special Interest (AESI)**

AESI will be defined per the version of the PSAP/MedDRA in effect at the time of DBR.

## Malignant Neoplasms

- Malignancies Excluding non-melanoma skin cancer (NMSC)
- Malignancies Including NMSC
  - Solid Tumour
  - Hematologic
  - Skin (All)
    - NMSC
    - Excluding NMSC
- Tumours of unspecified malignancy adjudicated as malignant per GSK

## Post-Infusion Systemic Reactions (PISR)

- PISR per Anaphylactic Reaction Customized MedDRA Query (CMQ) narrow search
- PISR per Anaphylactic Reaction CMQ broad search
- PISR per Anaphylactic Reaction CMQ algorithmic search
- Serious Anaphylaxis per Sampson Criteria per GSK adjudication
- Serious Acute PISR/Hypersensitivity Per GSK adjudication
  - Serious Acute PISR Excluding Hypersensitivity per GSK adjudication

#### **Adverse Events**

#### **Adverse Events of Special Interest (AESI)**

- Serious Acute Hypersensitivity Reactions per GSK adjudication
- Serious Delayed Acute Hypersensitivity Reactions per GSK adjudication
- Serious Delayed Non-Acute Hypersensitivity Reactions per GSK adjudication

## All Infections of Special Interest (Opportunistic Infections (OI), Herpes Zoster (HZ), Tuberculosis

## (TB), And Sepsis; All and Serious, separately)

- All opportunistic infections (OI) per GSK adjudication
- OI per GSK adjudication excluding Tuberculosis and Herpes Zoster
- Active Tuberculosis
  - Non-Opportunistic
  - Opportunistic
- Herpes Zoster
  - Non-Opportunistic
  - Opportunistic
    - Recurrent
    - Disseminated
- Sepsis

## <u>Depression (including mood disorders and anxiety)/suicide/self-injury (All and Serious, separately)</u>

- Depression (including mood disorders and anxiety) (excluding suicide and self-injury)
- Suicide/self-injury
- Serous suicide/self-injury per GSK adjudication
  - Suicidal Behaviour
    - Completed Suicide
  - Suicidal Ideation
  - Self-injurious Behaviour without Suicidal Intent
- Deaths

#### **Laboratory Parameters**

- If a laboratory value which is expected to have a numeric value for summary purposes, has a non-detectable level reported in the database, where the numeric value is missing, but typically a character value starting with '<x' or '>x' (or indicated as less than x or greater than x in the comment field) is present, the number of significant digits in the observed values will be used to determine how much to add or subtract in order to impute the corresponding numeric value.
  - Example 1: 2 Significant Digits = '< x ' becomes x 0.01
  - Example 2: 1 Significant Digit = '> x' becomes x + 0.1
- Example 3: 0 Significant Digits = '< x' becomes x − 1</li>

#### 13.6.5. Pharmacokinetic

#### Belimumab concentration

Assign zero to NQ values (Refer to GUI\_51487 for further details)

#### 13.6.6. Biomarker

## 13.6.6.1. Autoantibody, Complement, Immunoglobulins, and BLyS Protein

#### **Biomarker Categorical Definitions**

#### Anti-ds DNA

- Positive: ≥ 30 IU /mL
- Negative: < 30 IU /mL

#### ANA

- Positive: index ≥ 0.80
- Negative: index < 0.80

#### aCL status

- Positive: if any of the three isotypes IgG, IgA or IgM are above the lower limit of quantification
- Negative: if at least one isotype is non-missing and none of the isotypes are above the lower limit of quantification
- Missing: if all three isotypes are missing

## **BLyS** Protein

- Below LOQ: <0.02048 ng/mL</li>
- Above LOQ: ≥0.02048 ng/mL

#### C3

- Positive: < 90 mg/dL</li>
- Negative: ≥ 90 mg/dL
- Low: < 90 mg/dL</li>
- High: > 180 mg/dL

#### C4

- Positive: < 10 mg/dL</li>
- Negative: ≥ 10 mg/dL
- Low: < 10 mg/dL
- High: > 40 mg/dL

## Immunoglobulin G

- Low: < 6.94 g/L
- Normal/High: ≥ 6.94 g/L

## Immunoglobulin A

- Low: < 0.81 g/L
- Normal/High: ≥ 0.81 g/L

## Immunoglobulin M

- Low: < 0.48 g/L
- Normal/high: ≥ 0.48 g/L

#### 13.6.6.2. B-cell Subsets

## Flow Assays

B-cells can be assayed using 3 different flow panels (identification of the flow panel responsible for each record is stored in BIMETHCD in the data transfer): Not all assays
will have the full list of B-cells assessed, but data relating to CD19 B-cells are collected using all 3 assay methods, i.e. concentration of CD19 cells from the TBNK panel and CD19 event counts on the Plasma and Transitional panels (see detail in the table below).

Because the numbers of cells observed for the rare B-cell subsets are small, the concentration data cannot be adequately summarised in the units provided in the SI/SDTM data. Therefore, these subsets are normalized and converted to an appropriate unit of measurement, i.e. count/mL. To normalize a rare B-cell subset and convert to count/mL, the CD19+ B-cell event count from the same flow panel as the B-cell subset being converted is used in the derivation. For example, the CD19+ event count from the plasma flow panel is used to normalize B-cell subsets found in the plasma panel, whereas the CD19+ event count from the transitional panel is used when converting rare B-cell subsets from the transitional panel. The study RAP should detail which rare B-cell subsets will be normalized and converted.

#### Source data

Below are the important variables included in a source data transfer for the B-cells to be reported in this study.

| Flow Panel | Biomarker<br>testing<br>method<br>code | Biomarker<br>category<br>code<br>(BICATCD) <sup>1</sup> | Analyte name | Biomarker<br>test code<br>(BITESTCD) | Units of<br>Measurement<br>(BIORRESU) |
|---|---|---|---|---|---|
| TBNK | FLWTBNK | CD19 | CD19+ | CONC | GI/L |
| TBNK | FLWTBNK | CD19 | CD19+ | %LYMPH | % |
| PLASMA | FLWPLSM | CD19 | CD19+ | EVENTS | EVENTS |
| TRANSITIONAL | FLWTRANS | CD19 | CD19+ | EVENTS | EVENTS |
| PLASMA | FLWPLSM | CD20 | CD20+ | CONC | GI/L |
| PLASMA | FLWPLSM | CD20 | CD20+ | %CD19+ | % |
| PLASMA | FLWPLSM | CD20 | CD20+ | EVENTS | EVENTS |
| PLASMA | FLWPLSM | CDX136 | Naïve CD20+ CD27- | CONC | GI/L |
| PLASMA | FLWPLSM | CDX136 | Naïve CD20+ CD27- | %CD19+ | % |
| PLASMA | FLWPLSM | CDX136 | Naïve CD20+ CD27- | EVENTS | EVENTS |
| PLASMA | FLWPLSM | CDX137 | Memory CD20+ CD27+ | CONC | GI/L |
| PLASMA | FLWPLSM | CDX137 | Memory CD20+ CD27+ | %CD19+ | % |
| PLASMA | FLWPLSM | CDX137 | Memory CD20+ CD27+ | EVENTS | EVENTS |
| PLASMA | FLWPLSM | CDX141 | Activated CD20+ CD69+ | CONC | GI/L |
| PLASMA | FLWPLSM | CDX141 | Activated CD20+ CD69+ | %CD19+ | % |
| PLASMA | FLWPLSM | CDX143 | Plasma CD20- CD138+ | CONC | GI/L |
| PLASMA | FLWPLSM | CDX143 | Plasma CD20- CD138+ | %CD19+ | % |
| PLASMA | FLWPLSM | CDX143 | Plasma CD20- CD138+ | EVENTS | EVENTS |
| PLASMA | FLWPLSM | CDX145 | Plasmacytoid CD20+ CD138+ | CONC | GI/L |
| PLASMA | FLWPLSM | CDX145 | Plasmacytoid CD20+ CD138+ | %CD19+ | % |
| PLASMA | FLWPLSM | CDX145 | Plasmacytoid CD20+ CD138+ | EVENTS | EVENTS |
| PLASMA | FLWPLSM | CDX156 | SLE Subset CD27+CD38+CD19+ | CONC | GI/L |
| PLASMA | FLWPLSM | CDX156 | SLE Subset CD27+CD38+CD19+ | %CD19+ | % |
| PLASMA | FLWPLSM | CDX156 | SLE Subset CD27+CD38+CD19+ | EVENTS | EVENTS |

<sup>1</sup>Note: The SI data for Activated B-cells includes BICATCD=CDX141 for its concentration and %CD19 records, and CDX155 for its EVENTS record. For all other B-cell subsets, the BICATCD is the same for all 3 records.

#### B-cell unit conversions and Normalization of Rare B-cell Subsets

The Benlysta program standard is to report common B-cells (CD19, CD20, naïve, and memory) in counts per microliter (uL). Common B-cells are not normalized but they must be converted to uL for reporting. To convert values reported from GI/L (=  $10^9/L$ ) to count per uL (= cells/mm<sup>3</sup>), multiply the value by  $10^3$  or 1000.

Rare B-cell subsets are reported in counts per milliliter (mL). Rare B-cell subsets reported in GI/L will be converted to cells/ml using the following formula:

Note, the total B-cell (CD19+) concentration from the TBNK panel should be converted to count/uL prior to the normalization and conversion of the Rare B-cell subset.

Example: Normalization and conversion of Plasma CD20-CD138+ to count/mL

#### Given:

- Plasma CD20-CD138+ number of events = 16
- CD19+ number of events on Plasma panel = 10250
- CD19+ concentration on TBNK panel = 0.35 GI/L

#### Then:

Plasma CD20-CD138+ Normalized (count/mL) = 16 / 10250 \* (0.35\*1000) \* 1000 = 546.34 count/mL

#### Reporting B cell subsets

The table below includes variables, labels and details of derivations used in the reporting of the B-cell subsets for this study.

| | Lab Test<br>Code | Derivation for Normalization and / or Conversion |
|---|---|---|
| B-cell subset label for displays | (LBTESTCD) | of B-cell Subsets |
| Common B-cells | | |
| CD19 (/uL) | CD19 | May require conversion to /uL |
| CD20 (/uL) | CD20 | May require conversion to /uL |
| Naive CD19+CD20+CD27- (/uL) | CDX136 | May require conversion to /uL |
| Naive CD19+CD20+CD27- (%CD19) | CDX13619 | N/A |
| Memory CD19+CD20+CD27+ (/uL) | CDX137 | May require conversion to /uL |
| Memory CD19+CD20+CD27+ (%CD19) | CDX13719 | N/A |
| Rare B-cells | | |
| Activated CD19+CD20+CD69+ | CDX141N | CDX155 EVENTS, CD19 EVENTS from Plasma |
| Normalized (COUNT/mL) | | Panel and CD19 concentration from TBNK Panel |

| Plasma CD19+CD20-CD138+ | CDX143N | CDX143 EVENTS, CD19 EVENTS from Plasma |
|---|---|---|
| Normalized (COUNT/mL) | | Panel and CD19 concentration from TBNK Panel |
| Plasmacytoid CD19+CD20+CD138+ | CDX145N | CDX145 EVENTS, CD19 EVENTS from Plasma |
| Normalized (COUNT/mL) | | Panel and CD19 concentration from TBNK Panel |
| SLE Subset CD19+CD38b+CD27b+Lymph | CDX156N | CDX156 EVENTS, CD19 EVENTS from Plasma |
| Normalized (COUNT/mL) | | Panel and CD19 concentration from TBNK Panel |

# 13.7. Appendix 7: Reporting Standards for Missing Data

## 13.7.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | Subject study completion (i.e. as specified in the protocol) was defined as s |
| | <ul> <li>Treatment holiday group: completion of the 24-week treatment<br/>holiday period plus the belimumab re-introduction treatment period<br/>to Week 52.</li> </ul> |
| | <ul> <li>Control and long-term discontinuation groups: completion of all<br/>visits to Week 52.</li> </ul> |
| | For reporting purposes, withdrawal from the maintenance phase is defined in Section 13.6.2. |
| | Withdrawn subjects were not replaced in the study |
| | All available data from participants who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified. |
| | Withdrawal visits will be slotted as per Appendix 3: Assessment Windows or will be summarised as withdrawal visits. |

## 13.7.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument:</li> <li>These data will be indicated by the use of a "blank" in subject listing displays. Unless all data for a specific visit are missing in which case the data is excluded from the table.</li> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be missing data and should be displayed as such.</li> </ul> |
| Outliers | Any participants excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |
| LOCF | <ul> <li>In the LOCF dataset, missing values will be carried forward from the previous, non-missing available on-treatment assessment.</li> <li>For the TH group, LOCF will not be applied across the TH and RS phases.</li> </ul> |
| SLICC/ACR<br>Damage Index | <ul> <li>Missing data due to prohibited medication or study withdrawal will be imputed using LOCF</li> <li>For the TH group, LOCF will not be applied across the TH and RS phases.</li> </ul> |
| SELENA<br>SLEDAI, | <ul> <li>Missing data will be imputed using LOCF.</li> <li>For the TH group, LOCF will not be applied across the TH and RS phases.</li> </ul> |

| Element | Reporting Detail |
|---|---|
| Rebound, PGA | If an individual SELENA SLEDAI item data is missing at the first timepoint in the RS phase, the item will be considered not present. |
| Reduction in<br>Daily Prednisone<br>Dose | The Dropout (DO)/Prohibited Medication (PM)=Non-responder (NR) imputation will be applied. If a subject withdraws from the study and/or receives a protocol-prohibited medication prior to a scheduled visit, the subject will be considered a non-responder (i.e. no reduction in prednisone) for that and subsequent visits. |
| Average daily prednisone dose | Observed data will be used with no imputation. |
| Auto-antibodies,<br>immunoglobulins,<br>biomarkers, BLyS<br>protein | Observed data will be used with no imputation |
| Immunogenicity | Observed data will be used with no imputation. |

# 13.7.2.1. Handling of Missing and Partial Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in subject listing displays. |
| Adverse Events | <ul> <li>The eCRF allows for the possibility of partial dates (i.e., only month and year) to be recorded for AE start and end dates; that is, the day of the month may be missing. In such a case, the following conventions will be applied for calculating the time to onset and the duration of the event: <ul> <li>Missing Start Day: First of the month will be used unless this is before the start date of study treatment; in this case the Day 0 visit date (LTD and TH arms) or the study treatment start date (TC arm) will be used and hence the event is considered On-treatment as per Appendix 4: Study Phases and Treatment Emergent Adverse Events.</li> <li>Missing Stop Day: Last day of the month will be used, unless this is after the stop date of study treatment; in this case the study treatment stop date will be used.</li> </ul> </li> </ul> |
| | Completely missing start or end dates will remain missing, with no imputation applied. Consequently, time to onset and duration of such events will be missing. |
| Concomitant<br>Medications and<br>Medical History | <ul> <li>Medications with partial or missing start and/or stop dates will be assumed to be concomitant unless there is evidence through comparison of partial dates to suggest otherwise, for example if the day is missing, then the month and year will be compared to the month and year of the first dose date of study treatment and if the month and year are the same or later, then the medication will be considered concomitant.</li> </ul> |

# 13.7.3. Handling of Prohibited Medications, Withdrawals and Deaths

| Element | Reporting Detail |
|---|---|
| Time to SFI | Evaluated up to Week 52 |
| Flares | <ul> <li>If a subject takes a prohibited medication during the time period being<br/>analyzed, the subject will be considered as having a SFI flare at the start<br/>date of the prohibited medication.</li> </ul> |
| | If a subject withdraws from the study, the will be censored at last flare assessment date |
| | If a subject dies, censor at the date of death |
| Time to Renal | Evaluated up to Week 52 |
| Flare | If a subject withdraws from the study, the will be censored at last renal flare assessment date |
| | If a subject dies, censor at the date of death |
| Number of SFI<br>Flares | If a subject withdraws from the study, dies or takes a prohibited medication, the subject will be considered as having a SFI flare. |
| Number of days of daily prednisone dose ≥7.5 mg/day and/or increased by 25% | The Dropout (DO)/Prohibited Medication (PM)=Non-responder (NR) imputation will be applied. If a subject withdraws from the study and/or receives a protocol-prohibited medication, the subject will be considered to have met this endpoint criteria (i.e, dose ≥ 7.5 mg/day and/or increased by 25%) after the date of dropout or the date that the medication is started, whichever comes first, up until the visit date, and for those days in intervals for subsequent attended visits. Before this date, the evaluated endpoint will be assessed using available data. |
| Number of days<br>of daily<br>prednisone dose<br>≤7.5 mg/day<br>and/or<br>decreased by<br>25% | The Dropout (DO)/Prohibited Medication (PM)=Non-responder (NR) imputation will be applied. If a subject withdraws from the study and/or receives a protocol-prohibited medication, the subject will be considered a non-responder for this endpoint criteria (i.e., dose >7.5 mg/day and/or did not decreased by 25%) after the date of dropout or the date that the medication is started, whichever comes first, and for those days in intervals for subsequent attended visits. Before this date, the evaluated endpoint will be assessed using available data. |
| Reduction in<br>Daily<br>Prednisone<br>Dose | The Dropout (DO)/Prohibited Medication (PM)=Non-responder (NR) imputation will be applied. If a subject withdraws from the study and/or receives a protocol-prohibited medication prior to a scheduled visit, the subject will be considered a non-responder (i.e. no reduction in prednisone) for that and subsequent visits. |

# 13.8. Appendix 8: Values of Potential Clinical Importance

## 13.8.1. Laboratory Values

The following laboratory parameters are collected per the protocol.

| <u>Hematology</u> | <u>Urinalysis</u> | Modified Chem-20 |
|---|---|---|
| Total white blood cell count | Protein | Electrolytes: |
| Differential: | Glucose | Sodium |
| Absolute Neutrophils | Ketones | Potassium |
| Segmented Neutrophils | Occult blood | Magnesium |
| Band Neutrophils | Microscopic examination | Chloride |
| Myelocytes | including: | Carbon dioxide |
| Metamylocytes | WBC per hpf | Calcium adjusted for Albumin |
| Promyelocytes | RBC per hpf | Inorganic Phosphate |
| Lymphocytes | Dysmorphic RBC | F |
| Monocytes | Casts (specified by | Enzymes: |
| Eosinophils | type e.g., RBC, WBC) | SGOT (AST) |
| Basophils | Spot Urine (protein : creatinine | SGPT (ALT) |
| Hemoglobin | ratio) | Alkaline Phosphatase |
| Hematocrit | Urine Pregnancy | Gamma glutanyl transpeptidase (GGT) |
| Red blood cell (RBC) count | | Lactic dehydrogenase (LDH) |
| Platelet count | | 04 |
| Prothrombin time (PT) | | Other: |
| Partial thromboplastin time (PTT) | | Creatinine |
| | | Blood urea nitrogen (BUN) BUN/creatinine ratio |
| | | Bilirubin, total |
| | 1 | Protein, total Albumin |
| Biological Markers | | Uric acid |
| BLyS protein | | Glucose |
| Serum complement (C3 and C4) | | Hepatitis B Viral DNA PCR |
| B-cell subtypes | | Quantitative (HBV DNA) |
| ,, | | Estimated Creatinine Clearance/ GFR |
| <u>Immunoglobulins</u> | | (Cockroft-Gault) |
| Serum immunoglobulin isotypes: IgG, | gM, IgA | (Gockion-Gaun) |
| , | | Liver event follow-up assessments: |
| | | Hepatitis A IgM antibody |
| Immunogenicity | | HBsAg and hep B Core antibody (IgM) |
| | | Hepatitis C RNA |
| Autoantibodies | | Hepatitis delta antibody |
| ANA | | Cytomegalovirus IgM antibody |
| Anti-dsDNA | | Epstein-Barr viral capsid antigen IgM |
| aCL | | antibody |
| | | Hepatitis E IgM antibody |
| | | CPK |
| | | Anti-smooth muscle antibody |
| | | Type 1 anti-liver kidney microsomal |
| | | antibodies |
| | | PK |
| | | IgG |
| | | Fractionated bilirubin |
| | | Serum acetaminophen |

# 13.8.2. Adverse Event and Laboratory Value Severity Grade Tables

| HEMATOLOGY | GRADE 1<br>MILD | GRADE 2 MODERATE | GRADE 3 SEVERE | GRADE 4 POTENTIALLY LIFE-THREATENING |
|---|---|---|---|---|
| Hemoglobin | > 9.5 - 11.0 g/dL | > 8.0 – 9.5 g/dL | 6.5 - 8.0 g/dL | < 6.5 g/dL |
| Leukocytes | 3000-3999/mm3 | 2000-2999/mm3 | 1000-1999/mm3 | < 1000/mm3 |
| Absolute Neutrophil Count | 1500-1999/mm3 | 1000-1499/mm3 | 500-999/mm3 | < 500/mm3 |
| Platelets | 75,000 - | 50,000 – 74,999/mm3 | 25,000 - 49,999/mm3 | < 25,000/mm3 |
| | 99,999/mm3 | | | |
| Prothrombin Time (PT) | > 1.0-1.25 x ULN* | > 1.25-1.5 x ULN | > 1.5-3.0 x ULN | > 3.0 x ULN |
| Partial Thromboplastin Time (PTT) | > 1.0-1.66 x ULN | > 1.66-2.33 x ULN | > 2.33-3.0 x ULN | > 3.0 x ULN |
| Methemoglobin | 5.0-10.0 % | 10.1-15.0 % | 15.1-20.0 % | > 20% |
| | | | | (continued) |

<sup>1. \*</sup>ULN = Upper Limit of Normal

# **Adverse Event and Laboratory Value Severity Grade Tables (continued)**

| CARRIOVASCIII AR | GRADE 1 | GRADE 2 | GRADE 3 | GRADE 4 |
|---|---|---|---|---|
| CARDIOVASCULAR | MILD | MODERATE | SEVERE | POTENTIALLY LIFE-THREATENING |
| Cardiac Arrhythmia | - | Asymptomatic/transient;<br>dysrhythmia; no treatment req | Recurrent/persistent<br>dysrhythmia. Symptomatic;<br>treatment req | Unstable dysrhythmia hospitalization and treatment required |
| Hypotension | Transient orthostatic hypotension, no treatment | Symptoms correctable with oral fluid treatment | IV fluid req,<br>no hospitalization req | Hospitalization req |
| Hypertension | Transient, increase > 20 mm/Hg; no treatment | Recurrent; chronic increase > 20 mm/Hg, treatment req | Acute treatment req; out patient hospitalization possible | Hospitalization req |
| Pericarditis | Minimal effusion | Mild/moderate asymptomatic effusion, no treatment | Symptomatic effusion, pain, ECG changes | Tamponade OR pericardiocentesis OR surgery req |
| Hemorrhage, Blood Loss | - | Mildly symptomatic;<br>no treatment required | Gross blood loss OR<br>1-2 units transfused | Massive blood loss OR > 2 units transfused |
| Modified from DMID Adult Toxic | city Tables, 2001(continued) | | | <u> </u> |

# **Adverse Event and Laboratory Value Severity Grade Tables (continued)**

| | GRADE 1 | GRADE 2 | GRADE 3 | GRADE 4 |
|---|---|---|---|---|
| <u>CHEMISTRIES</u> | MILD | <u>MODERATE</u> | <u>SEVERE</u> | POTENTIALLY LIFE-THREATENING |
| Sodium | | | | L |
| Hyponatremia | 130-135 meq/L | 123-129 meq/L | 116-122 meq/L | < 116 meq/L |
| Hypernatremia | 146-150 meq/L | 151-157 meq/L | 158-165 meq/L | > 165 meq/L |
| Potassium | | | | |
| Hypokalemia | 3.0-3.4 meq/L | 2.5-2.9 meq/L | 2.0-2.4 meg/L | < 2.0 meq/L |
| Hyperkalemia | 5.6-6.0 meq/L | 6.1-6.5 meq/L | 6.6-7.0 meq/L | > 7.0 meq/L |
| Phosphate | | · | | |
| Hypophosphatemia | 2.0-2.4 mg/dL | 1.5-1.9 mg/dL | 1.0-1.4 mg/dL | < 1.0 mg/dL |
| Calcium- (Corrected For Albumin) | | | | • |
| Hypocalcemia | 7.8-8.4 mg/dL | 7.0-7.7 mg/dL | 6.1-6.9 mg/dL | < 6.1 mg/dL |
| Hypercalcemia | 10.6-11.5 mg/dL | 11.6-12.5 mg/dL | 12.6-13.5 mg/dL | >13.5 mg/dL |
| Magnesium | | | | |
| Hypomagnesemia | 1.2-1.4 meq/L | 0.9-1.1 meq/L | 0.6-0.8 meq/L | < 0.6 meq/L |
| Albumin | | | | |
| Hypoalbuminemia | 3.00-3.49 g/dL | 2.50-2.99 g/dL | 2.00-2.49 g/dL | < 2.00 g/dL |
| Bilirubin (Total) | | | | |
| Hyperbilirubinemia (Total) | > 1.0-1.5 x ULN | > 1.5-2.5 x ULN | > 2.5-5 x ULN | > 5 x ULN |
| Glucose | | | | |
| Hypoglycemia | 55-64 mg/dL | 40-54 mg/dL | 30-39 mg/dL | < 30 mg/dL |
| Hyperglycemia | 116-160 mg/dL | 161-250 mg/dL | 251-500 mg/dL | > 500 mg/dL |
| (nonfasting & no prior diabetes) | | | | |
| Triglycerides | 151-399 mg/dL | 400-750 mg/dL | 751-1200 mg/dL | > 1200 mg/dL |
| Creatinine | > 1.0-1.5 x ULN | > 1.5-3.0 x ULN | > 3.0-6.0 x ULN | > 6.0 x ULN |
| | | | | (continued) |

# **Adverse Event and Laboratory Value Severity Grade Tables (continued)**

| | GRADE 1 | GRADE 2 | GRADE 3 | GRADE 4 |
|---|---|---|---|---|
| CHEMISTRIES (continued) | MILD | <u>MODERATE</u> | <u>SEVERE</u> | POTENTIALLY LIFE-THREATENING |
| Uric Acid | | | | I |
| Hyperuricemia | 7.5-10.0 mg/dL | 10.1-12.0 mg/dL | 12.1-15.0 mg/dL | > 15.0 mg/dL |
| Liver Transferases (AST, ALT, and GGT) | 1.25-2.5 x ULN | > 2.5-5.0 x ULN | > 5.0-10.0 x ULN | > 10.0 x ULN |
| Alkaline Phosphatase | 1.25-2.5 x ULN | > 2.5-5.0 x ULN | > 5.0-10.0 x ULN | > 10.0 x ULN |
| Pancreatic Enzymes | | • | • | • |
| Amylase | > 1.0-1.5 x ULN | > 1.5-2.0 x ULN | > 2.0-5.0 x ULN | > 5.0 x ULN |
| Pancreatic amylase | > 1.0-1.5 x ULN | > 1.5-2.0 x ULN | > 2.0-5.0 x ULN | > 5.0 x ULN |
| Lipase | > 1.0-1.5 x ULN | > 1.5-2.0 x ULN | > 2.0-5.0 x ULN | > 5.0 x ULN |
| Hypoglobulinemia (IgG)* | 550-700 mg/dL | 400-549 mg/dL | 250-399 mg/dL | < 250 mg/dL |
| | | | | (continued) |

<sup>1. \*</sup>Eibl , 1995; Goldfarb, 2001; Yamini, 2001.

# **Adverse Event and Laboratory Value Severity Grade Tables (continued)**

| | GRADE 1 | GRADE 2 | GRADE 3 | GRADE 4 |
|---|---|---|---|---|
| GASTROINTESTINAL | MILD | MODERATE | SEVERE | POTENTIALLY LIFE-THREATENING |
| Nausea | Mild OR transient;<br>reasonable intake<br>maintained | Mod discomfort OR intake decreased for < 3 days | Severe discomfort OR minimal intake for ≥ 3 days | Hospitalization required |
| Vomiting | Mild OR transient;<br>2-3 episodes/day OR<br>mild vomiting lasting<br>< 1 week | Mod OR persistent;<br>4-5 episodes per day;<br>OR vomiting lasting<br>≥ 1 week | Severe vomiting of all foods/fluids in 24 hours OR orthostatic hypotension OR IV treatment req | Hypotensive shock OR hospitalization required for IV treatment req |
| Diarrhea | Mild or transient; 3-4 loose stools per day OR mild diarrhea lasting < 1 week | Mod OR persistent;<br>5-7 loose stools per day<br>or diarrhea lasting<br>≥ 1 week | Bloody diarrhea;<br>OR orthostatic hypotension<br>OR > 7 loose stools/day<br>OR IV treatment req | Hypotensive shock OR hospitalization req |
| Oral Discomfort/Dysphagia | Mild discomfort, no difficulty swallowing | Difficulty swallowing but able to eat and drink | Unable to swallow solids | Unable to drink fluids;<br>IV fluids req |
| Constipation | Mild | Moderate | Severe | Distention with vomiting (continued) |

# **Adverse Event and Laboratory Value Severity Grade Tables (continued)**

| | GRADE 1 | GRADE 2 | GRADE 3 | GRADE 4 |
|---|---|---|---|---|
| RESPIRATORY | MILD | MODERATE | <u>SEVERE</u> | POTENTIALLY LIFE-THREATENING |
| Cough<br>(for aerosol studies) | Transient; no treatment | Treatment associated cough; inhaled bronchodilator | Uncontrolled cough;<br>systemic treatment req | |
| Bronchospasm Acute | Transient; no treatment;<br>FEV1 70% to<br>< 80%<br>(or peak flow) | treatment req; normalizes with<br>bronchodilator;<br>FEV1 50% to < 70%<br>(or peak flow) | No Normalization<br>with bronchodilator;<br>FEV 25% to < 50%<br>(or peak flow), retractions | Cyanosis; FEV1 < 25%<br>(or peak flow) OR intubated |
| Dyspnea | Dyspnea on exertion | Dyspnea with normal activity | Dyspnea at rest | Dyspnea requiring O2 therapy |

# **Adverse Event and Laboratory Value Severity Grade Tables (continued)**

| | GRADE 1 | GRADE 2 | GRADE 3 | GRADE 4 |
|---|---|---|---|---|
| <u>URINALYSIS</u> | MILD | MODERATE | SEVERE | POTENTIALLY LIFE-THREATENING |
| Proteinuria | | | | |
| Dispstick | | | | |
| Protein | 1 + | 2-3 + | 4 + | Nephrotic syndrome |
| Spot Urine: | 0.2-1.0 | > 1.0-2.0 | > 2.0-3.5 | > 3.5 |
| Protein:Creatinine | 0.2 1.0 | 1.0 2.0 | 2.0 0.0 | 0.0 |
| Ratio mg/mg | | | | |
| 24 Hour Urine: | 200 mg - 1g loss/day | > 1-2 g loss/day | > 2-3.5 g loss/day | Nephrotic syndrome |
| Protein | | | | OR > 3.5 g loss/day |
| Hematuria | Microscopic only | Gross, No clots | Gross plus clots OR | Obstructive OR transfusion required |
| | > 3 to < 10 RBC/hpf | ≥ 10 RBC/hpf | RBC casts | · · |
| | | • | | (continued) |
| RBC = red blood cell; hp | f = high power field. | | | |
| | | | | Modified from DMID Adult Toxicity Tables, 2001 |

# **Adverse Event and Laboratory Value Severity Grade Tables (continued)**

| MISCELLANEOUS | GRADE 1 MILD | GRADE 2 MODERATE | GRADE 3 SEVERE | GRADE 4 POTENTIALLY LIFE-THREATENING |
|---|---|---|---|---|
| Fever (oral > 12 hours) | 37.7-38.5°C or<br>100.0-101.5°F | 38.6-39.5°C OR<br>101.6-102.9°F | 39.6-40.5°C OR<br>103-105°F | > 40.5°C OR > 105°F |
| Headache | Mild; No treatment req | Mod; or non-narcotic analgesia treatment | Severe; OR responds to initial narcotic treatment | Intractable; OR requiring repeated narcotic treatment |
| Allergic Reaction | Pruritus without rash | Localized urticaria | Generalized urticaria angioedema | Anaphylaxis |

| MISCELLANEOUS | GRADE 1<br>MILD | GRADE 2 MODERATE | GRADE 3 SEVERE | GRADE 4 POTENTIALLY LIFE-THREATENING |
|---|---|---|---|---|
| Cutaneous/Rash/ Dermatitis | Erythema, pruritus rash<br>OR dry desquamation | Diffuse maculopapular<br>OR dry desquamation | Vesiculation OR moist desquamation ulceration | ANY ONE: mucous membrane involvement, suspected Stevens-Johnson (TEN), erythema multiforme, necrosis req surgery, exfoliative dermatitis |
| Local Reaction (secondary to parenteral treatment- not vaccination or skin test) | Erythema | Induration < 10 mm OR inflammation OR phlebitis | Induration > 10 mm OR ulceration | Necrosis of skin |
| Fatigue | Normal activity<br>Reduced < 25% | Normal activity<br>Reduced 25-50% | Normal activity reduced > 50%; cannot work | Unable to care for self |
| | l | | | (continued) |

# **Adverse Event and Laboratory Value Severity Grade Tables (continued)**

| | GRADE 1 | GRADE 2 | GRADE 3 | GRADE 4 |
|---|---|---|---|---|
| NEUROLOGIC | MILD | MODERATE | SEVERE | POTENTIALLY LIFE-THREATENING |
| Neuro-cerebellar | Slight incoordination OR dysdiadochokinesia | Intention tremor OR<br>dysmetria OR slurred speech<br>OR nystagmus | Ataxia requiring assistance to walk or arm incoordination interfering with ADLs | Unable to stand |
| Neuro-psych/ mood | | none | Severe mood changes requires medical intervention | Acute psychosis requiring hospitalization |
| Paresthesia (burning, tingling, etc) | Mild discomfort;<br>no treatment needed | Mod discomfort<br>non-narcotic analgesia req | Severe discomfort; OR narcotic analgesia req with symptomatic improvement | Incapacitating; OR not responsive to narcotic analgesia |
| Neuro-motor | Mild weakness in muscle<br>of feet but<br>able to walk and/or mild<br>increase or decrease in<br>reflexes | Mod weakness in feet (unable to walk on heels and/or toes), mild weakness in hands, still able to do most hand tasks and/or loss of previously present reflex or development of hyperreflexia and/or unable to do deep knee bends due to weakness | Marked distal weakness (unable to dorsiflex toes or foot drop), and mod proximal weakness ie, in hands interfering with ADLs and/or requiring assistance to walk and/or unable to rise from chair unassisted | Confined to bed or wheelchair because of muscle weakness |
| Neuro-sensory | Mild impairment<br>sensations,<br>(ie, vibratory, pinprick,<br>hot/cold in great toes) in<br>focal area or symmetrical<br>distribution | Mod impairment mod de-sensation, (ie, of vibratory, pinprick, hot/cold to ankles) and/or joint position or mild impairment that is not symmetrical. | Severe impairment (dec or loss of sensation to knees or wrists) or loss of sensation of at least mod degree in multiple different body areas (ie, upper and lower extremities) | Sensory loss involves limbs and trunk |
| | | | | (concluded) |

### 13.9. Appendix 9: Adverse Events of Special Interest

The primary source for rules governing identification, adjudication, and reporting of Adverse Events of Special Interest is the Program Safety Analysis Plan (PSAP). AESI are defined using preferred terms from the current version of MedDRA. The intent is to update these definitions semi-annually using the newest MedDRA version. Preferred terms used in the current and prior versions of MedDRA can be found in IMMS at the following path /Study File/GSK1550188/ Project/Meta Analysis/PSAP/AESI 201.csv.

### 13.9.1. Malignant neoplasms

Malignant neoplasms are identified using the sub-SMQs of Malignant or unspecified tumours (20000091), malignancy related conditions (20000092), haematological malignant tumours (20000227), non-haematological malignant tumours (20000228), haematological tumours of unspecified malignancy (20000229) and non-haematological tumours of unspecified malignancy (20000230) under the current version of MedDRA. The sub-SMQ of Malignant or unspecified tumours contains two further subcategories: "Malignant Tumours" and "Tumours of unspecified malignancy." Tumours of unspecified malignancy will be reviewed by GSK and identified as malignant or non-malignant for reporting.

Malignancies other than those in the "Tumours of unspecified malignancy" category will be categorized as hematologic, skin, or solid, based on a CMQ developed by the MAH. In addition, the following customizations have been made since MedDRA v19.1:

- The term "Paraneoplastic glomerulonephritis" has been removed from the SMQ as it is a complication of malignancy.
- The term "Mismatch repair cancer syndrome" has been added as a tumour of unspecified malignancy
- The term "Malignant meningioma metastatic" has been added as a solid tumor type.
- The term "Marginal zone lymphoma recurrent" has been added as a hematological tumor type.
- The term "Skin neoplasm bleeding" has been added as a tumour of unspecified malignancy.
- The term "Astroblastoma" has been added as a solid tumour type.
- The term "Epstein Barr virus positive mucocutaneous ulcer" has been added as a hematological tumour type.
- The term "Langerhans cell sarcoma" has been added as a solid tumour type.
- The term "Naevoid melanoma" has been added as a skin tumour type.
- The term "Nasopharyngeal cancer metastatic" has been added as a solid tumour type.
- The term "Phospaturic mesenchymal tumour" has been added as a solid tumour type.
- The term "Primary gastrointestinal follicular lymphoma" has been added as a hematological tumour type.

- The term "Squamous cell breast carcinoma" has been added as a solid tumour type.
- The term "Transformation to acute myeloid leukaemia" has been added as a hematological tumour type.
- The term "FIP1L1/PDGFR alpha fusion kinase positive" has been added as a hematological tumour type.
- The term "Gleason grading score" has been added as a solid tumour type.
- The term "Oncotype test" has been added as a solid tumour type.
- The term "Intestinal metastasis" has been added as an unspecified tumour type.
- The term "Maternal cancer in pregnancy" has been added as an unspecified tumour type.
- The term "Microsatellite instability cancer" has been added as an unspecified tumour type.
- The term "Pulmonary tumour thrombotic microangiopathy" has been added as an unspecified tumour type.
- The term "Tumour cavitation" has been added as an unspecified tumour type.
- The term "Malignant urinary tract obstruction" has been added as a solid tumour type.

Non-melanoma skin cancer (NMSC) will be categorized using a CMQ developed by the Marketing authorization holder (MAH)

Note beginning with MedDRA v20.0 in 2017, there will be two new sub-SMQs of Hematological Malignancies. These do not result in any changes to how malignant neoplasms are identified.

## 13.9.2. Post-infusion systemic reactions

Post-infusion systemic reactions will be identified using a customization of the Anaphylactic Reaction SMQ (20000021). This SMQ includes a broad list of preferred terms including symptoms of systemic injection/infusion reactions and hypersensitivity reactions and anaphylaxis. For the Anaphylactic Reaction query, 4 categories of preferred terms are considered, including a set of core anaphylactic terms (Category A), upper airway/respiratory terms (Category B), angioedema/urticaria/pruritus/flush terms (Category C), and cardiovascular/hypotension terms (Category D).

The customizations of the SMQ involve terms in Categories A, B and C. Category A has been modified to include the following additional terms: "Infusion-related reaction", "Drug hypersensitivity", "Hypersensitivity", and "Urticarial vasculitis". Category B has been modified to include the following additional terms: "Oropharyngeal oedema" and "Pharyngeal oedema". Category C has been modified to include the following additional term: "Fixed eruption". GSK has also removed three terms that are not relevant for an analysis of hypersensitivity reactions to belimumab ("Anaphylactic transfusion reaction", "Dialysis membrane reaction", and "First use syndrome"). Anaphylactic transfusion reaction is an adverse event associated with a blood transfusion, not related to study

medication. First use syndrome and dialysis membrane reaction are associated with adverse events related to kidney transplants and dialysis, not related to study medication.

#### **Algorithmic Search Criteria**

The post-infusion systemic reactions per Anaphylactic Reaction SMQ algorithmic search are defined as follows:

Subjects must have the following associated with the same infusion/injection:

- a. at least 1 AE coding to a Category A preferred term or
- b. 2 AEs, 1 coding to a Category B preferred term and the other coding to a Category C preferred term *or*
- c. 2 AEs, 1 coding to a Category D preferred term and the other coding to either a Category B preferred term or to a Category C preferred term.

For the algorithmic search, if any event at a given infusion/injection meets the definition under criteria a, b or c, then all events in Categories A, B, C and D associated with that injection/infusion will be considered AESI.

For CSR reporting, all post-infusion systemic reaction AESIs defined via narrow, broad, or algorithmic search, the AEs need to have occurred on the day of an infusion/injection or within 3 days after an infusion/injection. See Section 13.3.4 for the definition of the 3-day assessment window. GSK will review all serious events identified via the broad search occurring within 21 days after an infusion/injection, and adjudicate these events as post-infusion systemic reactions or hypersensitivity reactions per the criteria in Section 13.9.10.2. Adverse events with partial or missing start dates will be included unless there is evidence through comparison of partial dates to suggest otherwise.

#### Sampson Criteria

Sampson et al define anaphylaxis as a severe, potentially fatal, systemic allergic reaction that occurs suddenly after contact with an allergy-causing substance. In addition, one of the following 3 criteria must be met: (1) acute onset of illness with involvement of skin or mucosal tissue, accompanied with either respiratory compromise, reduced blood pressure, or hypotension-related symptoms of end-organ dysfunction (2) reduced blood pressure associated with a known allergen or (3) two or more of the following that occur rapidly after exposure to an allergen: a) involvement of skin-mucosal tissue b) respiratory compromise c) reduced blood pressure d) persistent GI symptoms.

With the exception of GI symptoms, all symptoms required to assess anaphylaxis per Sampson criteria would be identified by Broad Anaphylaxis SMQ or the Anaphylactic Reaction SMQ algorithmic. Therefore, any events falling under the below criteria will be adjudicated by GSK prior to database release to determine if serious anaphylaxis per Sampson criteria is met.

Possible cases of serious anaphylaxis per Sampson criteria will be identified as follows:

a. Any Infusion/Injection-related Reaction per Anaphylactic Reaction SMQ broad

- search SAE which occurs on the day of an injection.
- b. Any AE or SAE in the "Gastrointestinal disorders" SOC that occurs on the day that criterion in a) above is met.
- c. Any anaphylaxis and hypersensitivity reactions per Anaphylactic Reaction SMQ algorithmic search SAE which occurs on the day of an infusion/injection.

#### 13.9.3. Infections

The infections of special interest are described below.

#### 13.9.3.1. Opportunistic Infections

Opportunistic infections will be identified using a broad CMQ developed by the MAH. Any events falling under these preferred terms will be adjudicated by GSK prior to database release to determine if criteria are met for an opportunistic infection, per the criteria in Section 13.9.10.3.

#### 13.9.4. Mycobacterium Tuberculosis

Tuberculosis events will be identified using a CMQ developed by the MAH. Any events falling under these preferred terms will be adjudicated by GSK prior to database release to determine if criteria are met for an opportunistic infection (Section 13.9.10.3).

#### 13.9.5. Herpes Zoster

Herpes Zoster events will be identified using a CMQ developed by the MAH. Additional manual adjudication by GSK prior to database release will identify events that are recurrent or disseminated (Section 13.9.10.3).

#### 13.9.6. Pneumonia

Pneumonia events will be identified using a CMQ developed by the MAH. Pneumonia events will not be reported separately, but are being flagged in the event further evaluation is necessary.

#### 13.9.7. Sepsis

Sepsis events will be identified using a CMQ developed by the MAH.

### 13.9.8. Depression/suicide/self-injury

#### 13.9.8.1. Depression (excluding suicide and self-injury)

Depression events will be identified using a CMQ including the preferred terms from the depression (excluding suicide and self injury) SMQ (20000035) plus additional terms added by the MAH.

#### 13.9.8.2. Suicide and Self-Injury

Suicide and self-injury events will be identified using the SMQ (20000035) preferred terms.

#### 13.9.9. Fatalities

All fatalities will be identified in the clinical database and subsequently adjudicated by the GSK SRT into a general category of death (Section 13.9.10.5).

Post-study fatalities that are captured in ARGUS prior to CSR approval, but are not captured in the clinical database, will be described within the CSR text but cannot be included in statistical post-text displays.

## 13.9.10. GSK SRT Adjudication of Adverse Events of Special Interest

Adverse events of special interest (AESI) are identified per the preferred terms and other criteria described in Section 13.9. The following AESI are adjudicated at the subject level by the GSK SRT during regular SRT meetings or during quarterly adjudication. The adjudication occurs prior to database release and is performed for reporting purposes, per the criteria described below.

Assignment of adjudication flags in the clinical database will occur as part of the quarterly SRT review process. In addition, as part of individual study close-out procedures, the adjudications should be finalized as follows:

- Just preceding data base release (DBR), allowing time to send queries or update the eCRF/database as necessary prior to DBR.
- After DBR to provide final confirmation of adjudications and ensure there are no new AESI or relevant data changes to adjudicated events since the pre-DBR adjudication. This would be a requirement for declaring data a freeze (DBF).

#### 13.9.10.1. Malignancies

All malignancies identified via the preferred terms will be reviewed by GSK SRT. The classification of malignancies as solid tumor, hematological, and skin will be reviewed against the verbatim term to confirm an appropriate and accurate preferred term has been assigned, or to recommend follow-up with the investigator for additional specificity on the verbatim term. In addition, malignancies that are flagged more than once, e.g., based on a term for both a diagnostic procedure and a diagnosis, will be adjudicated as one event.

Tumors of unspecified malignancy, as identified via preferred terms, will be reviewed clinically by the GSK SRT for reporting. In general, non-serious events in the tumours of unspecified malignancy with insufficient information will be categorized as not malignant. Serious adverse events with insufficient information will be categorized as either not malignant or malignant based on the type of tumor and likelihood the tumor type is malignant (e.g., thyroid nodules are common in SLE patients and are generally not

malignant; tumor types with higher likelihood for malignancy would be assumed to be malignant).

#### 13.9.10.2. Serious hypersensitivity and post-infusion systemic reactions

Before the data base is released, GSK SRT will review all serious cases identified from the Broad Anaphylaxis SMQ as described in Section 13.9, applying clinical judgment to determine if the preferred terms are indicative of a hypersensitivity or infusion/injection reaction. Time to onset after an infusion/injection and details provided in the clinical narratives with respect to the nature and likely cause of the events are taken into consideration. Time to onset within 24 hours is generally applied to post infusion/injection reactions. The GSK SRT adjudicates serious hypersensitivity reactions into a category based primarily on time to onset: acute (onset  $\leq$  1 day), delayed acute (onset 2-3 days), or delayed, non-acute (onset 4-21 days). In addition to time to onset, description of associated symptoms is taken into account for this categorization.

In addition, possible cases of serious anaphylaxis per Sampson criteria will be identified per the criteria in Section 13.9. Any events falling under these criteria will be adjudicated by GSK prior to database release to determine if serious anaphylaxis per Sampson criteria is met.

#### 13.9.10.3. Potential opportunistic infections

Opportunistic infections (OIs) will be identified using a list of preferred terms, designed to cast a wide net for events potentially indicative of an opportunistic infection. Any identified events will be adjudicated by the GSK SRT prior to database release to determine if criteria are met for an opportunistic infection. Targeted follow-up is sought for events with insufficient information. In general, potential OIs that are non-serious with insufficient information to adjudicate will be considered non-opportunistic. Potential OI SAEs with insufficient information to adjudicate will be considered opportunistic. See below for a list of agreed upon pathogens and infections considered to be opportunistic for the purpose of adjudication.

#### **Pathogens and Infections Considered Opportunistic:**

- Acinetobacter infection
- Aspergillosis
- Blastomycosis, extrapulmonary
- Candidiasis of esophagus, bronchi, trachea or lungs
- Coccidioidomycosis, disseminated or extrapulmonary
- Cryptococcosis, extrapulmonary
- Cryptosporidiosis infection, chronic intestinal (greater than 1 month duration)
- CMV disease other than liver, spleen, or nodes
- Herpes simplex bronchitis, pneumonitis, or esophagitis
- Herpes Zoster (adjudication details are below)
- Histoplasmosis disseminated or extrapulmonary
- Human polyomavirus infection
- Isosporiasis, chronic intestinal (greater than one month duration)

- Listeriosis
- Mycobacterium avium complex or M. Kansasii, disseminated or extrapulmonary
- Nocardiosis
- Other non-tuberculous mycobacterium (NTM) infections (other species or unidentified species), disseminated or extrapulmonary\*
- Polyomavirus (JC virus or BK virus) associated nephropathy (including PML)
- Pneumocystis jiroveci infection
- Toxoplasmosis of brain
- \* Extra pulmonary NTM infections are generally considered an OI unless the affected extra pulmonary area followed a wound or trauma.

In addition, GSK SRT will review all SAEs, including those coded under preferred terms not in the preferred term definition, and utilizing the supplemental/narrative information, will adjudicate the SAEs as OI if warranted based on medical judgment.

#### Other Infections of Interest but not generally considered opportunistic:

• Mycobacterium tuberculosis (adjudication details are below)

#### **Herpes Zoster**

Herpes Zoster events will be identified per preferred terms. Adjudication by GSK SRT will identify events that are recurrent or disseminated. Herpes Zoster is considered disseminated if there is involvement of other organs other than the skin or if skin lesions (1) cross the midline of the body or (2) are in non-adjacent dermatomes or (3) are located in more than three adjacent dermatomes. Herpes zoster is considered an opportunistic infection if it is adjudicated as recurrent or disseminated. However, there may be some uncommon occurrences of a herpes zoster case that is adjudicated as an OI but is neither recurrent or disseminated.

#### **Mycobacterium Tuberculosis**

Tuberculosis (TB) cases are reviewed by the GSK SRT to determine if a case is an OI. The following principles are applied: Pulmonary TB in an endemic area is not considered an OI. Pulmonary TB in a non-endemic area would be considered an OI unless the subject had close contact with a person infected with TB. Extra pulmonary TB is generally considered an OI unless the affected extra pulmonary area followed a wound or trauma.

#### 13.9.10.4. Suicide/self-injury

Suicide and self-injury SAEs will be identified using the preferred terms and subsequently adjudicated into the following categories:

| Adjudicated Category |
|--------------------------------------------------|
| Suicidal Behaviour |
| Completed Suicide |
| Suicidal Ideation |
| Self-Injurious Behaviour without Suicidal Intent |

In addition, GSK SRT will review all SAEs, including those coded under preferred terms not in the definition, and utilizing the supplemental/narrative information, will adjudicate the SAEs as suicide/self-injury if warranted based on medical judgment.

#### 13.9.10.5. Fatalities

All fatalities will be identified in the clinical database and subsequently adjudicated by the GSK SRT into a general category of death.

All fatalities will be adjudicated into one of the following categories:

| <b>Adjudicated Category of Death</b> |
|--------------------------------------|
| SLE-Related |
| Infectious |
| Vascular |
| Gastrointestinal |
| Respiratory |
| Malignancy |
| Hypersensitivity |
| Suicide |
| Surgical Complication |
| Unknown |
| Hematologic |
| Trauma |

Additional 'categories of death' may be added in the future should a fatality not clearly fit into one of the 'categories' listed above. The 'categories' will not change unless agreed upon by the GSK SRT.

# 13.10. Appendix 10: Abbreviations & Trade Marks

## 13.10.1. Abbreviations

| Abbreviation | Description |
|---|---|
| ADaM | Analysis Data Model |
| aCL | Anti-cardiolipin Antibody |
| ACR | American College of Rheumatology |
| AE | Adverse Event |
| AESI | AEs of Special Interest |
| Anti-dsDNA | Anti-double-stranded DNA |
| ANA | Anti-nuclear Antibody |
| ATC | Anatomical Therapeutic Chemical |
| BMI | Body mass index |
| BUN | Blood urea nitrogen |
| CDISC | Clinical Data Interchange Standards Consortium |
| C3 / C4 | Complement 3 / Complement 4 |
| CI | Confidence Interval |
| CNS | Central Nervous System |
| CRF | Case Report Form |
| CS | Clinical Statistics |
| CSR | Clinical Study Report |
| eCRF | Electronic Case Report Form |
| DO | Dropout |
| DOB | Date of Birth |
| DP DOB | Decimal Places |
| DQE | |
| eCRF | Data Quality Evaluation Report Electronic Case Report Form |
| GFR | Glomerular Filtration Rate |
| GSK | GlaxoSmithKline |
| GUI | Guidance |
| hpf<br>ICH | High-power Field International Conference on Harmonisation |
| IDSL | Integrated Data Standards Library |
| IgA, G, M | Immunoglobulin A, G, M |
| IM | Intramuscular |
| IMMS | International Modules Management System |
| ITT | Intention-to-treat |
| IV | Intravenous |
| LLN | Lower Limit of Normal |
| LOCF | Last Observation Carried Forward |
| LOQ | Limit of Quantification |
| LTD | Long-term discontinuation |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MHE | Mental Health Enhanced Score |
| NMSC | Non-melanoma skin cancer |
| NR | Non-responder |
| Ol | Opportunistic Infections |
| PCI | Potential Clinical Importance |
| PD | Pharmacodynamic |

| Abbreviation | Description |
|--------------|-----------------------------------------------------|
| PDMP | Protocol Deviation Management Plan |
| PGA | Physician's Global Disease Assessment |
| PK | Pharmacokinetic |
| PM | Prohibited medication |
| PopPK | Population Pharmacokinetic |
| PSAP | Program Safety Analysis Plan |
| PT | Preferred Term/Prothrombin Time |
| PTT | Partial thromboplastin Time |
| QC | Quality Control |
| RAP | Reporting and Analysis Plan |
| RAMOS | Randomization & Medication Ordering System |
| RBC | Red blood cell |
| RS | Re-start Phase |
| SAC | Statistical Analysis Complete |
| SAE | Serious Adverse Event |
| SC | Subcutaneous |
| SD | Standard deviation |
| SDTM | Study Data Tabulation Model |
| SE | Standard error |
| SELENA | Safety of Estrogen in Lupus National Assessment |
| SI | System independent |
| SFI | SLE Flare Index |
| SLE | Systemic Lupus Erythematosus |
| SLEDAI | Systemic Lupus Erythematosus Disease Activity Index |
| SLICC | Systemic Lupus International Collaborating Clinics |
| SMQ | Standardized MedDRA Query |
| SoC | Standard of Care |
| SOC | System Organ Class |
| SOP | Standard Operation Procedure |
| SS | SELENA SLEDAI |
| TC | Treatment Control |
| TH | Treatment Holiday |
| TLFs | Tables, Listings, and Figures |
| TX | Treatment |
| ULN | Upper Limit of Normal |
| uPCR | Urine Protein: Creatinine Ratio. |
| VAS | Visual Analogue Scale |
| WOCF | Worst Observation Carried Forward |

## 13.10.2. Trademarks

| Trademarks of the GlaxoSmithKline<br>Group of Companies |
|---------------------------------------------------------|
| BENLYSTA |
| BLyS |

Trademarks not owned by the GlaxoSmithKline Group of Companies

# 13.11. Appendix 11: List of Data Displays

# 13.11.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------|-------------|-------------|
| Study Population | 1.1 to 1.17 | 1.1 to 1.1 |
| Efficacy | 2.1 to 2.12 | 2.1 to 2.3 |
| Safety | 3.1 to 3.52 | 3.1 to 3.6 |
| Pharmacokinetic | 4.1 to 4.1 | 4.1 to 4.2 |
| Biomarker | 5.1 to 5.23 | 5.1 to 5.10 |
| Section | Listings | |
| ICH Listings | 1 to 39 | |
| Other Listings | 40 to | o 51 |

## 13.11.2. Deliverables

| Priority | Description |
|----------|-----------------------------------|
| Н | Included in Headline Data Package |

# 13.11.3. Study Population Tables

| Study P | opulation Table | s | | |
|---|---|---|---|---|
| No. | Population | Title | Programming Notes | Priority<br>Headline Results<br>denoted by H |
| Subject | Disposition | | | |
| 1.1. | ITT | Subject Enrollment | | |
| 1.2. | ITT | Enrolment by Country and Site | EudraCT/Clinical Operations | |
| 1.3. | Screened | Study Populations | IDSL | |
| 1.4. | Screened | Screening Status and Reasons for Failing Screening | Journal Requirements | |
| 1.5. | ITT | Subject Disposition for the Subject Conclusion Record (52-Week Treatment Phase) | ICH E3, FDAAA, EudraCT | |
| 1.6. | ITT | Subject Disposition for the Subject Conclusion Record (Maintenance Phase) | ICH E3, FDAAA, EudraCT | |
| 1.7. | ITT | Time to Withdrawal from the Study | Benlysta Standard | |
| 1.8. | ITT | Subject Disposition at Each Study Epoch | ICH E3 | |
| Protoco | l Deviation | | | • |
| 1.9. | ITT | Subjects with Important Protocol Deviations | ICH E3 | |
| Demogr | aphic and Base | line Characteristics | | |
| 1.10. | ITT | Demographic and Baseline Characteristics | ICH E3, FDAAA, EudraCT | Н |
| 1.11. | ITT | Age Ranges | EudraCT | |
| 1.12. | ITT | Race and Racial Combination Details | ICH E3, FDA, FDAAA, EudraCT | |
| Current a | and Prior Medical | History | | |
| 1.13. | ITT | General Medical History | ICH E3 | |

| Study P | Study Population Tables | | | |
|---|---|---|---|---|
| No. | Population | Title | Programming Notes | Priority<br>Headline Results<br>denoted by H |
| Baseline | Baseline Disease Activity and SLE Medication Use | | | |
| 1.14. | ITT | Baseline Disease Activity | Benlysta Standard | Н |
| 1.15. | ITT | SELENA SLEDAI Organ and Item Involvement at Baseline | Benlysta Standard | Н |
| 1.16. | ITT | Allowable SLE Medication Usage at Baseline | Benlysta Standard | |
| 1.17. | ITT | Steroid, Anti-malarial and Immunosuppressant Use at Baseline | Benlysta Standard | |

# 13.11.4. Study Population Figures

| Study Pop | Study Population: Figure | | | |
|---|---|---|---|---|
| No. | No. Population Title Programming Notes Priority | | | |
| Time to W | Time to Withdrawal | | | |
| 1.1 | ITT | Time to Withdrawal | Study Population | Н |

# 13.11.5. Efficacy Tables

| Efficacy | : Tables | | | |
|---|---|---|---|---|
| No. | Population | Title | Programming Notes | Priority<br>Headline Results<br>denoted by H |
| Flares | | | | |
| 2.1. | ITT | Time to First SFI Flare to Week 52 | Primary endpoint | Н |
| 2.2. | ITT | SFI Flares per Subject-year from Day 0 to Week 52 | Secondary endpoint | |
| 2.3. | ITT | Time to First SFI Severe Flare to Week 52 | Secondary endpoint | Н |
| 2.4. | ITT | Time to First Renal Flare to Week 52 | Exploratory endpoint | Н |
| 2.5. | ITT | Time to First Renal Flare to Week 52 [1] Among Subjects with Baseline Proteinuria >0.5g/24hr Equivalent | Exploratory endpoint | |
| Rebound | d and SELENA- | SLEDAI | | |
| 2.6. | ITT | SELENA SLEDAI Rebound (LOCF) (52-Week Treatment Phase) | Secondary endpoint | Н |
| 2.7. | ITT | SELENA SLEDAI Change from Baseline (LOCF) (52-Week Treatment Phase) | Secondary endpoint | |
| PGA | | | | |
| 2.8. | ITT | PGA Change from Baseline (52-Week Treatment Phase) | Other/exploratory endpoint | |
| Predniso | one | | | |
| 2.9. | ITT | Number of Days of Daily Prednisone Dose >=7.5 mg/day and/or Increased by 25% | Secondary endpoint | |
| 2.10. | ITT | Number of Days of Daily Prednisone Dose <=7.5 mg/day and/or Decreased by 25% | Secondary endpoint | |

| Efficacy | Efficacy: Tables | | | |
|---|---|---|---|---|
| No. | Population | Title | Programming Notes | Priority<br>Headline Results<br>denoted by H |
| 2.11. | ITT | Prednisone Percent Change from Baseline (52-Week Treatment Phase) | Other/exploratory endpoint | |
| 2.12. | ITT | Prednisone Reduced to <= 7.5 mg/day by Visit (DO/TF=NR) among Subjects with Baseline Prednisone Dose > 7.5 mg/day (52-Week Treatment Phase) | Other/exploratory endpoint | |

# 13.11.6. Efficacy Figures

| Efficacy | Efficacy: Figures | | | |
|---|---|---|---|---|
| No. | Population | Title | Programming Notes | Priority |
| Flares | | | , | |
| 2.1. | ITT | Time to First SFI Flare to Week 52 | Primary endpoint | Н |
| 2.2. | ITT | Time to First Severe SFI Flare to Week 52 | Secondary endpoint | Н |
| Reboun | Rebound and SELENA-SLEDAI | | | |
| 2.3. | ITT | SELENA SLEDAI Change from Baseline by Visit (LOCF) (52-Week Treatment Phase) | Secondary endpoint | |

# 13.11.7. Safety Tables

| Safety: | Safety: Tables | | | |
|---|---|---|---|---|
| No. | Population | Title | Programming Notes | Priority<br>Headline Results<br>Denoted by H |
| Conco | mitant Medicati | ons | | |
| 3.1. | ITT | Concomitant Medications by ATC Level 1 and ATC Level 4 Term for the 52-Week Treatment Phase | ICH E3 | |
| Study A | Agent Exposur | e | | |
| 3.2. | ITT | Study Agent Exposure (52-Week Treatment Phase) | ICH E3 | |
| SLICC | | | | |
| 3.3. | ITT | SLICC/ACR Damage Index Change from Baseline (52-Week Treatment Phase) | Other/exploratory endpoint | |
| Advers | e Events | | | |
| 3.4. | ITT | Adverse Events (52-Week Treatment Phase) | Benlysta standard | Н |
| 3.5. | ITT | Adverse Events by SOC (52-Week Treatment Phase) | Benlysta standard | |
| 3.6. | ITT | Serious Adverse Events by SOC (52-Week Treatment Phase) | Benlysta standard | |
| 3.7. | ITT | Study Agent Related Adverse Events by SOC (52-Week Treatment Phase) | Benlysta standard | |
| 3.8. | ITT | Adverse Events Resulting in Study Agent Discontinuation by SOC (52-Week Treatment Phase) | Benlysta standard | |

| Safety: | Tables | | | |
|---|---|---|---|---|
| No. | Population | Title | Programming Notes | Priority<br>Headline Results<br>Denoted by H |
| 3.9. | ITT | Adverse Events by SOC and PT (52-Week Treatment Phase) | ICH E3 | Н |
| 3.10. | ITT | Serious Adverse Events by SOC and PT (52-Week Treatment Phase) | Benlysta Standard | Н |
| 3.11. | ITT | Study Agent Related Adverse Events by SOC and PT (52-Week Treatment Phase) | ICH E3 | |
| 3.12. | ITT | Adverse Events Resulting in Study Agent Discontinuation by SOC and PT (52-Week Treatment Phase) | IDSL | Н |
| 3.13. | ITT | Adverse Events by PT (52-Week Treatment Phase) | Benlysta Standard | |
| 3.14. | ITT | Serious Adverse Events by PT (52-Week Treatment Phase) | Benlysta Standard | |
| 3.15. | ITT | Study Agent Related Adverse Events by PT (52-Week Treatment Phase) | Benlysta Standard | |
| 3.16. | ITT | Adverse Events Resulting in Study Agent Discontinuation by PT (52-Week Treatment Phase) | Benlysta Standard | |
| 3.17. | ITT | Common (>5%) Non-Serious Adverse Events by SOC and PT (52-Week Treatment Phase) (Number of Subjects and Occurrences) | FDAAA, EudraCT | |
| 3.18. | ITT | Serious Adverse Events by SOC and PT (52-Week Treatment Phase) (Number of Participants and Occurrences) | FDAAA, EudraCT | Н |
| 3.19. | ITT | Adverse Events by SOC and PT and Maximum Severity (52-Week Treatment Phase) | IDSL | |

| Safety: | Tables | | | |
|---|---|---|---|---|
| No. | Population | Title | Programming Notes | Priority<br>Headline Results<br>Denoted by H |
| 3.20. | ITT | Relationship Between System Organ Class and Verbatim Text (52-Week Treatment Phase) | IDSL | |
| 3.21. | ITT | Adverse Events of Special Interest by Category (52-Week Treatment Phase) | Benlysta Standard | Н |
| 3.22. | ITT | Adverse Events of Special Interest by Category and Infusion for Treatment Holiday Group Re-Start Phase | Benlysta Standard | |
| Labora | tory Parameter | s | | |
| 3.23. | ITT | Laboratory Results by Visit: Hematology (52-Week Treatment Phase | | |
| 3.24. | ITT | Laboratory Results by Visit: Liver Function (52-Week Treatment Phase) | | |
| 3.25. | ITT | Laboratory Results by Visit: Electrolytes (52-Week Treatment Phase) | | |
| 3.26. | ITT | Laboratory Results by Visit: Other Chemistries (52-Week Treatment Phase) | | |
| 3.27. | ITT | Laboratory Results by Visit: Urinalysis (52-Week Treatment Phase) | | |
| 3.28. | ITT | Laboratory Results by Visit: Immunoglobulins (52-Week Treatment Phase) | | |
| 3.29. | ITT | Worst Laboratory Toxicity Grade: Hematology (52-Week Treatment Phase) | ICH E3 | |

| Safety: | Safety: Tables | | | |
|---|---|---|---|---|
| No. | Population | Title | Programming Notes | Priority<br>Headline Results<br>Denoted by H |
| 3.30. | ITT | Worst Laboratory Toxicity Grade: Liver Function (52-Week Treatment Phase) | ICH E3 | |
| 3.31. | ITT | Worst Laboratory Toxicity Grade: Electrolytes (52-Week Treatment Phase) | ICH E3 | |
| 3.32. | ITT | Worst Laboratory Toxicity Grade: Other Chemistries (52-Week Treatment Phase) | ICH E3 | |
| 3.33. | ITT | Worst Laboratory Toxicity Grade: Urinalysis (52-Week Treatment Phase) | ICH E3 | |
| 3.34. | ITT | Worst Laboratory Toxicity Grade: Immunoglobulins (52-Week Treatment Phase) | ICH E3 | |
| 3.35. | ITT | Laboratory Toxicity Grade Worsening of at Least 2 Grades from Baseline: Hematology (52-Week Treatment Phase) | Benlysta Standard | |
| 3.36. | ITT | Laboratory Toxicity Grade Worsening of at Least 2 Grades from Baseline: Liver Function (52-Week Treatment Phase) | Benlysta Standard | |
| 3.37. | ITT | Laboratory Toxicity Grade Worsening of at Least 2 Grades from Baseline: Electrolytes (52-Week Treatment Phase) | Benlysta Standard | |
| 3.38. | ITT | Laboratory Toxicity Grade Worsening of at Least 2 Grades from Baseline: Other Chemistries (52-Week Treatment Phase) | Benlysta Standard | |
| 3.39. | ITT | Laboratory Toxicity Grade Worsening of at Least 2 Grades from Baseline: Urinalysis (52-Week Treatment Phase) | Benlysta Standard | |
| 3.40. | ITT | Laboratory Toxicity Grade Worsening of at Least 2 Grades from Baseline: Immunoglobulins (52-Week Treatment Phase) | Benlysta Standard | |
| 3.41. | ITT | Laboratory Reference Range Shifts from Baseline by Visit:<br>Hematology (52-Week Treatment Phase) | Benlysta Standard | |

| Safety: Tables | | | | |
|---|---|---|---|---|
| No. | Population | Title | Programming Notes | Priority Headline Results Denoted by H |
| 3.42. | ITT | Laboratory Reference Range Shifts from Baseline by Visit: Liver Function (52-Week Treatment Phase) | Benlysta Standard | |
| 3.43. | ITT | Laboratory Reference Range Shifts from Baseline by Visit: Electrolytes (52-Week Treatment Phase) | Benlysta Standard | |
| 3.44. | ITT | Laboratory Reference Range Shifts from Baseline by Visit: Other Chemistries (52-Week Treatment Phase) | Benlysta Standard | |
| 3.45. | ITT | Laboratory Reference Range Shifts from Baseline by Visit: Urinalysis (52-Week Treatment Phase) | Benlysta Standard | |
| 3.46. | ITT | Laboratory Reference Range Shifts from Baseline by Visit: Immunoglobulins (52-Week Treatment Phase) | Benlysta Standard | |
| lmmun | oglobulins | | | |
| 3.47. | ITT | Immunoglobulin Levels below the Lower Limit of Normal (LLN) by Visit (52-Week Treatment Phase) | Benlysta Standard | |
| 3.48. | ITT | Immunoglobulins below the Lower Limit of Normal (LLN) at each Visit among Subjects with Immunoglobulins >= LLN at Baseline (52-Week Treatment Phase) | Benlysta Standard | |
| 3.49. | ITT | Immunoglobulins above the Lower Limit of Normal (LLN) at each Visit (52-Week Treatment Phase) | Benlysta Standard | |
| 3.50. | ITT | Immunoglobulins above the Lower Limit of Normal (LLN) at each Visit among Subjects with Immunoglobulins <= LLN at Baseline (52-Week Treatment Phase) | Benlysta Standard | |
| lmmun | ogenicity | | | |
| 3.51. | ITT | Immunogenic Response by Visit (52-Week Treatment Phase) | Benlysta Standard | |
| Safety: | Safety: Tables | | | | | |
|---|---|---|---|---|--|--|
| No. | Population | Title | Programming Notes | Priority<br>Headline Results<br>Denoted by H | | |
| Vital Signature | Vital Signs | | | | | |
| 3.52. | ITT | Vital Signs Change from Baseline by Visit (Observed) (52-Week Treatment Phase) | ICH E3 | | | |

## 13.11.8. Safety Figures

| Safety: | Safety: Figures | | | |
|---|---|---|---|---|
| No. | Population | Title | Programming Notes | Priority |
| Labora | tory | | | |
| 3.1. | ITT | Laboratory Results by Visit: Hematology (52-Week Treatment Phase) | | |
| 3.2. | ITT | Laboratory Results by Visit: Liver Function (52-Week Treatment Phase) | | |
| 3.3. | ITT | Laboratory Results by Visit: Electrolytes (52-Week Treatment Phase) | | |
| 3.4. | ITT | Laboratory Results by Visit: Other Chemistries (52-Week Treatment Phase) | | |
| 3.5. | ITT | Laboratory Results by Visit: Other Chemistries (52-Week Treatment Phase) | | |
| 3.6. | ITT | Laboratory Results by Visit: Immunoglobulins (52-Week Treatment Phase) | | |

### 13.11.9. Pharmacokinetic Tables

| Pharma | Pharmacokinetic: Tables | |
|---|---|---|
| No. | No. Population Title Programming Notes Priority | |
| Belimui | Belimumab Concentrations | |
| 4.1. | PK | Belimumab Concentrations (ug/ml) |

## 13.11.10. Pharmacokinetic Figures

| Pharma | Pharmacokinetic: Figures | | | |
|---|---|---|---|---|
| No. | Population | Title | Programming Notes | Priority |
| Belimu | mab Concentra | ations | , | |
| 4.1. | PK | Median Belimumab Concentrations (ug/mL): 52-Week Treatment Phase | | |
| 4.2. | PK | Geometic Mean Belimumab Concentrations (ug/mL): 52-Week Treatment Phase | | |

### 13.11.11. Biomarker Tables

| Biomar | Biomarker Tables | | | |
|---|---|---|---|---|
| No. | Population | Title | Programming Notes | Priority |
| Autoan | tibodies | 1 | | |
| 5.1. | ITT | Autoantibody Levels Change from Baseline by Visit (Observed) (52-Week Treatment Phase) | | |
| 5.2. | ITT | Autoantibody Levels Percent Change from Baseline by Visit (Observed) (52-Week Treatment Phase) | | |
| 5.3. | ITT | Autoantibody Levels Change from Baseline by Visit among Subjects Positive at Baseline (Observed) (52-Week Treatment Phase) | | |

| Biomar | Biomarker Tables | | | |
|---|---|---|---|---|
| No. | Population | Title | Programming Notes | Priority |
| 5.4. | ITT | Autoantibody Levels Percent Change from Baseline by Visit among Subjects Positive at Baseline (Observed) (52-Week Treatment Phase) | | |
| 5.5. | ITT | Autoantibody Levels Shift from Baseline by Visit (Observed) (52-Week Treatment Phase) | | |
| Comple | ement | | | |
| 5.6. | ITT | Complement Levels Change from Baseline by Visit (Observed) (52-Week Treatment Phase) | | |
| 5.7. | ITT | Complement Levels Percent Change from Baseline by Visit (Observed) (52-Week Treatment Phase) | | |
| 5.8. | ITT | Complement Levels Change from Baseline by Visit among Subjects Low at Baseline (Observed) (52-Week Treatment Phase) | | |
| 5.9. | ITT | Complement Levels Percent Change from Baseline by Visit among Subjects Low at Baseline (Observed) (52-Week Treatment Phase) | | |
| 5.10. | ITT | Complement Levels Shift from Baseline by Visit (Observed) (52-Week Treatment Phase) | | |

| Biomai | Biomarker Tables | | | |
|---|---|---|---|---|
| No. | Population | Title | Programming Notes | Priority |
| Immun | mmunoglobulins | | | |
| 5.11. | ITT | Immunoglobulins Change from Baseline by Visit (Observed) (52-Week Treatment Phase) | | |
| 5.12. | ITT | Immunoglobulins Percent Change from Baseline by Visit (Observed) (52-Week Treatment Phase) | | |
| 5.13. | ITT | Immunoglobulins Change from Baseline by Visit among Subjects Low at Baseline (Observed) (52-Week Treatment Phase) | | |
| 5.14. | ITT | Immunoglobulins Percent Change from Baseline by Visit among Subjects Low at Baseline (Observed) (52-Week Treatment Phase) | | |
| 5.15. | ITT | Immunoglobulin Levels Shift from Baseline by Visit (Observed) (52-Week Treatment Phase) | | |
| B-cells | | | | |
| 5.16. | ITT | B-cells Change from Baseline by Visit (Observed) (52-Week Treatment Phase) | | |
| 5.17. | ITT | B-cells Percent Change from Baseline by Visit (Observed) (52-Week Treatment Phase) | | |
| 5.18. | ITT | B-cells Change from Baseline by Visit (Observed) (52-Week Treatment Phase) | | |
| 5.19. | ITT | B-cells Percent Change from Baseline by Visit (Observed) (52-Week Treatment Phase) | | |
| 5.20. | ITT | B-cells Change from Week 24 by Visit (Observed) (Maintenance Phase) | | |

| Biomar | Biomarker Tables | | | |
|---|---|---|---|---|
| No. | Population | Title | Programming Notes | Priority |
| 5.21. | ITT | B-cells Percent Change from Week 24 by Visit (Observed) (Maintenance Phase) | | |
| BLyS P | rotein | | | |
| 5.22. | ITT | BLyS ProteinChange from Baseline by Visit (Observed) (52-Week Treatment Phase) | | |
| 5.23. | ITT | BLyS Protein Percent Change from Baseline by Visit (Observed) (52-Week Treatment Phase) | | |

# 13.11.12. Biomarker Figures

| Biomarker Fi | Biomarker Figures | | | |
|---|---|---|---|---|
| No. | Population | Title | Programming Notes | Priority |
| Autoantibodi | es | | | |
| 5.1. | ITT | Autoantibody Levels Percent Change from Baseline by Visit (52-Week Treatment Phase) | | |
| 5.2. | ITT | Autoantibody Levels Percent Change from Baseline by Visit among Subjects Positive at Baseline (52-Week Treatment Phase) | | |
| Complement | | | | |
| 5.3. | ITT | Complement Levels Percent Change from Baseline by Visit (52-Week Treatment Phase) | | |
| 5.4. | ITT | Complement Levels Percent Change from Baseline by Visit among Subjects Positive at Baseline (52-Week Treatment Phase) | | |

| Biomarker Fi | Biomarker Figures | | | |
|---|---|---|---|---|
| No. | Population | Title | Programming Notes | Priority |
| Immunoglobu | ılins | | | |
| 5.5. | ITT | Immunoglobulin Levels Percent Change from Baseline by Visit (52-Week Treatment Phase) | | |
| 5.6. | ITT | Immunoglobulin Levels Percent Change from Baseline by Visit among Subjects Positive at Baseline (52-Week Treatment Phase) | | |
| BLyS Protein | | | | |
| 5.7. | ITT | BLyS Protein Percent Change from Baseline by Visit (52-Week Treatment Phase) | | |
| B cell Subset | S | | | |
| 5.8. | ITT | B Cell Percent Change from Baseline by Visit (52-Week Treatment Phase) | | |
| 5.9. | | B Cell Percent Change from Week 24 by Visit (52-Week Treatment Phase) | | |
| 5.10. | ITT | B Cell Absolute Values by Visit and Subject for Subjects who Enter the Maintenance Phase | | |

## 13.11.13. ICH Listings

| ICH: Li | ICH: Listings | | | |
|---|---|---|---|---|
| No. | Population | Title | Programming Notes | Priority |
| Subjec | Subject Disposition | | | |
| 1. | Screened | Reasons for Screen Failure | Journal requirements | |
| 2. | Screened | Re-Screened Subjects | | |
| 3. | ITT | Subject Disposition and Population Status | ICH E3 | |
| 4. | ITT | Previous Trial History | ICH E3 | |
| 5. | ITT | Reasons for Study Withdrawal | ICH E3 | |
| Protoc | ol Deviations | | | |
| 6. | Screened | Subjects with Inclusion/Exclusion Criteria Deviations | ICH E3 | |
| 7. | Screened | Important Protocol Deviations | ICH E3 | |
| Demog | graphic and Ba | seline Characteristics | | |
| 8. | ITT | Demographic and Baseline Characteristics | ICH E3 | |
| 9. | ITT | General Medical History | ICH E3 | |
| 10. | ITT | Subjects Who Took Prohibited Medications | Study specific | |
| Prior a | nd Concomita | nt Medications | | |
| 11. | ITT | Concomitant Medications | ICH E3 | |
| Expos | Exposure and Treatment Compliance | | | |
| 12. | 12. ITT Study Agent Administration ICH E3 | | | |
| Advers | se Events | | | |
| 13. | ITT | All Adverse Events | ICH E3 | |

| ICH: Li | ICH: Listings | | | |
|---|---|---|---|---|
| No. | Population | Title | Programming Notes | Priority |
| 14. | ITT | Subject Numbers for Individual Adverse Events | ICH E3 | |
| 15. | ITT | Relationship Between Adverse Event System Organ Classes, Preferred Terms, and Verbatim Text | IDSL | |
| Seriou | s and Other Si | gnificant Adverse Events | | |
| 16. | ITT | Serious Adverse Events | Study specific/ ICH E3 (other significant events) | |
| 17. | ITT | Deaths | ICH E3 | |
| 18. | ITT | Non-Fatal Serious Adverse Events | ICH E3 | |
| 19. | ITT | Study Treatment Related Adverse Events | Study specific/ ICH E3 (other significant events) | |
| 20. | ITT | Adverse Events Resulting in Study Treatment Discontinuation | ICH E3 | |
| 21. | ITT | Pre-treatment Adverse Events | Study specific/ ICH E3 (other significant events) | |
| 22. | ITT | Adverse Events of Special Interest | Study specific/ ICH E3 (other significant events) | |
| 23. | ITT | Malignancy Adverse Events of Special Interest | Study specific/ ICH E3 (other significant events) | |
| 24. | ITT | Reasons for Considering as a Serious Adverse Event | ICH E3 | |
| 25. | ITT | Infusion Related Systemic Reactions | Study specific | |
| 26. | ITT | Concomitant Procedures/Surgery | Study specific | |
| Vital S | Vital Signs | | | |
| 27. | 27. ITT Vital Signs IDSL | | | |
| All Lab | oratory | | | |
| 28. | ITT | Laboratory Results: Hematology | | |

| ICH: Listings | | | | |
|---|---|---|---|---|
| No. | Population | Title | Programming Notes | Priority |
| 29. | ITT | Laboratory Results: Liver Function | | |
| 30. | ITT | Laboratory Results: Electrolytes | | |
| 31. | ITT | Laboratory Results: Other Chemistries | | |
| 32. | ITT | Laboratory Results: Urinalysis | | |
| 33. | ITT | Laboratory Results: Immunoglobulins | | |
| 34. | ITT | Grade 3 or Grade 4 Laboratory Toxicity Results: Hematology | | |
| 35. | ITT | Grade 3 or Grade 4 Laboratory Toxicity Results: Liver Function | | |
| 36. | ITT | Grade 3 or Grade 4 Laboratory Toxicity Results: Electrolytes | | |
| 37. | ITT | Grade 3 or Grade 4 Laboratory Toxicity Results: Other Chemistries | | |
| 38. | ITT | Grade 3 or Grade 4 Laboratory Toxicity Results: Urinalysis | | |
| 39. | ITT | Grade 3 or Grade 4 Laboratory Toxicity Results: Immunoglobulins | | |
| Hepato | biliary (Liver) | | | |
| 40. | ITT | Liver Monitoring Stopping Event Reporting | | |
| 41. | ITT | Medical Conditions for Participants with Liver Stopping Events | | |
| 42. | ITT | Substance Use for Participants with Liver Stopping Events | | |

# 13.11.14. Non-ICH Listings

| Non-ICH: Listings | | | | |
|---|---|---|---|---|
| No. | Population | Title | Programming Notes | Priority |
| Efficacy Endpoints | | | | |
| 43. | ITT | SFI Flares | Study specific | |
| 44. | ITT | SELENA-SLEDAI Analysis Results | Study specific | |
| 45. | ITT | Physician's Global Assessment (PGA) Analysis Results | Study specific | |
| 46. | ITT | Average Daily Prednisone Dose | Study specific | |
| Immunogenicity | | | | |
| 47. | ITT | Immunogenicity Results | Study specific | |
| SLICC | | | | |
| 48. | ITT | SLICC/ACR Damage Index Analysis Results | Study specific | |
| Belimumab PK Concentration | | | | |
| 49. | PK | Serum Belimumab PK Concentration-Time Data | Study specific | |
| Biomarkers | | | | |
| 50. | ITT | Autoantibody and Complement Results | Study specific | |
| 51. | ITT | B Cell Results | Study specific | |

## 13.12. Appendix 12: Example Mock Shells for Data Displays

Data Display Specification will be made available on Request